CLINICAL TRIAL: NCT00866619
Title: Efficacy of GSK Biologicals' Candidate Malaria Vaccine (257049) Against Malaria Disease Caused by P. Falciparum Infection in Infants and Children in Africa
Brief Title: Efficacy of GSK Biologicals' Candidate Malaria Vaccine 257049 Against Malaria Disease in Infants and Children in Africa
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: The PATH Malaria Vaccine Initiative (MVI) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 110021; 2012-005716-26 (EudraCT Number)
Record Dates: First submitted 2009-03-19; First posted 2009-03-20 (Estimated); Results first posted 2019-10-09 (Actual); Last update posted 2019-10-09 (Actual); Status verified 2019-09

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria | interventions — RTS malaria vaccine; serogroup C meningococcal conjugate vaccine; halofantrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (4):
- GSK257049 [5-17M] Group (Experimental): Male or female children between and including 5 to 17 months of age [5-17M], who received a 3-dose primary vaccination course of the GSK257049 malaria vaccine, according to a 0-1-2 Month schedule, followed by either a booster dose of the same GSK257049 vaccine or a dose of Menjugate vaccine, at Month 20. Both vaccines have been administered intramuscularly into the left deltoid.
  Interventions: Biological: Malaria Vaccine 257049; Biological: Meningococcal C Conjugate Vaccine
- GSK257049 [6-12W] Group (Experimental): Male or female children between and including 6 to 12 weeks of age [6-12W], who received a 3-dose primary vaccination course of the GSK257049 malaria vaccine co-administered with Polio Sabin and Tritanrix HepB/Hib vaccines, according to a 0-1-2 Month schedule, followed by either a booster dose of the GSK257049 and Polio Sabin vaccines or a booster dose of Menjugate and Polio Sabin vaccines, at Month 20. All vaccines have been administered intramuscularly in the interolateral left thigh (GSK257049 vaccine); left deltoid (GSK257049 booster dose); left thigh for children under 1 year and left deltoid for children above 1 year of age (Menjugate vaccine); anterolateral right thigh (Tritanrix HepB/Hib vaccine), except for the Polio Sabin vaccine, which has been given orally.
  Interventions: Biological: Malaria Vaccine 257049; Biological: Meningococcal C Conjugate Vaccine; Biological: TritanrixHepB/Hib; Biological: Polio Sabin Oral Polio Vaccine (GSK)
- VeroRab Comparator [5-17M] Group (Active Comparator): Male or female children between and including 5 to 17 months of age [5-17M], who received a 3-dose primary vaccination course of the VeroRab vaccine, according to a 0-1-2 Month schedule, followed by a booster dose of Menjugate vaccine, at Month 20. Both vaccines have been administered intramuscularly into the left deltoid.
  Interventions: Biological: Meningococcal C Conjugate Vaccine; Biological: Cell-culture rabies vaccine
- Menjugate Comparator [6-12W] Group (Experimental): Male or female children between and including 6 to 12 weeks of age [6-12W], who received a 3-dose primary vaccination course of Menjugate vaccine co-administered with Polio Sabin and Tritanrix HepB/Hib vaccines, according to a 0-1-2 Month schedule, followed by a booster dose of Menjugate and Polio Sabin vaccines, at Month 12. All vaccines have been administered intramuscularly in the left thigh for children under 1 year and left deltoid for children above 1 year of age (Menjugate vaccine); anterolateral right thigh (Tritanrix HepB/Hib vaccine), except for the Polio Sabin vaccine, which has been given orally.
  Interventions: Biological: Meningococcal C Conjugate Vaccine; Biological: TritanrixHepB/Hib; Biological: Polio Sabin Oral Polio Vaccine (GSK)

INTERVENTIONS:
Biological: Malaria Vaccine 257049 — administered intramuscularly into the left deltoid.
  Arms: GSK257049 [5-17M] Group; GSK257049 [6-12W] Group
Biological: Meningococcal C Conjugate Vaccine — administered intramuscularly into the left deltoid.
  Other Names: Menjugate
Biological: Cell-culture rabies vaccine — administered intramuscularly into the left deltoid.
  Other Names: VeroRab
  Arms: VeroRab Comparator [5-17M] Group
Biological: TritanrixHepB/Hib — administered intramuscularly into the left deltoid.
  Arms: GSK257049 [6-12W] Group; Menjugate Comparator [6-12W] Group
Biological: Polio Sabin Oral Polio Vaccine (GSK) — administered orally.
  Arms: GSK257049 [6-12W] Group; Menjugate Comparator [6-12W] Group

SUMMARY:
The purpose of this observer-blind study is to gather key efficacy, safety, and immunogenicity information on GSK's candidate malaria vaccine in infants and children.

DETAILED DESCRIPTION:
The protocol posting document has been updated due to a protocol amendment dated 23 January 2012. An analysis time point has been added at Month 20. No changes have been made to the protocol endpoints or statistical methods but protocol endpoints will be analysed on data collected up to Month 20 once these data are available. The rationale is to have the full scope of protocol defined efficacy and safety endpoints related to a primary schedule without booster in both age categories followed up for 20 months earlier than at the initially planned study end time point (Visit 34 or Month 32 time point).

The protocol posting document was updated due to a protocol amendment dated 10 December 2010 to extend the study until December 2013 for all enrolled subjects (interval: Nov 2013-Jan 2014). Including the extension, the mean follow-up time for subjects from 5-17 months will be during 49 months post dose 1 (range: 41-55), while for subjects from 6-12 weeks, it will be during 41 months post dose 1 (range: 32-48). This study is double-blind during the first part and single-blind during the extension part. An analysis will be conducted at the end of the extension including an evaluation of safety and efficacy against clinical malaria, severe malaria and prevalent parasitemia.

The protocol posting document has been updated following the posting of results of the study (January 2015): The study remained double-blind until the end of the extension phase, and the analyses of Month 32 (initial end of study now becoming end of the first part of the study or primary study phase) and of the extension phase were conducted together.

ELIGIBILITY:
Inclusion Criteria:

All subjects must satisfy the following criteria at study entry:

* A male or female child of:5-17 months (inclusive) of age at time of first vaccination,or between 6-12 weeks of age at time of first vaccination and NOT have already received a dose of vaccine against diphtheria, tetanus or pertussis or Hemophilus influenzae type B and must be > 28 days of age at screening.
* Signed informed consent or thumb-printed and witnessed informed consent obtained from the parent(s)/guardian(s) of the child.
* Subjects who the investigator believes that their parents/guardians can and will comply with the requirements of the protocol.

All subjects must satisfy the following criteria at the start of the extension phase:

* Subjects who were enrolled and who received at least one vaccine dose in the primary trial phase.
* Subjects who were present for Visit 35 on or before 30 September 2013.
* Subjects who the investigator believes that their parents/guardians can and will comply with the requirements of the protocol (e.g. return for follow-up visits) should be enrolled in the study.

Exclusion Criteria:

The following criteria should be checked at the time of study entry. If any apply, the subject must not be included in the study:

* Acute disease at the time of enrollment.
* Acute or chronic, clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality.
* Anemia associated with clinical signs or symptoms of decompensation or hemoglobin ≥ 5.0 g/dL.
* Major congenital defects.
* History of allergic reactions, significant IgE-mediated events or anaphylaxis to previous immunizations.
* Children with a past history of a neurological disorder or atypical febrile seizure.
* Children with malnutrition requiring hospital admission.
* Children currently meeting the criteria for HIV disease of Stage III or Stage IV severity as defined by the World Health Organization.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to a drug or vaccine that is not licensed for that indication with the exception of studies with the objective of improving the drug treatment or clinical management of severe malaria disease.
* Use of a drug or vaccine that is not approved for that indication other than the study vaccines within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Previous participation in any other malaria vaccine trial.
* Receipt of a vaccine within the preceding 7 days.
* Any other findings that the investigator feels would increase the risk of having an adverse outcome from participation in the trial.
* Any other findings that the investigator feels would result in data collected being incomplete or of poor quality

Ages: 6 Weeks to 17 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 15459 (Actual)
Dates: Start 2009-03-27 (Actual); Primary Completion 2011-03-01 (Actual); Study Completion 2014-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (10):
- GSK Investigational Site, Ouagadougou, Burkina Faso
- GSK Investigational Site, Lambaréné, Gabon
- Ghana (2):
  - GSK Investigational Site, Kintampo
  - GSK Investigational Site, Kumasi
- Kenya (2):
  - GSK Investigational Site, Kilifi
  - GSK Investigational Site, Kisumu
- GSK Investigational Site, Lilongwe, Malawi
- GSK Investigational Site, Maputo, Mozambique
- Tanzania (2):
  - GSK Investigational Site, Dar es Salaam
  - GSK Investigational Site, Tanga

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

REFERENCES:
- [Background] RTS,S Clinical Trials Partnership; Agnandji ST, Lell B, Fernandes JF, Abossolo BP, Methogo BG, Kabwende AL, Adegnika AA, Mordmuller B, Issifou S, Kremsner PG, Sacarlal J, Aide P, Lanaspa M, Aponte JJ, Machevo S, Acacio S, Bulo H, Sigauque B, Macete E, Alonso P, Abdulla S, Salim N, Minja R, Mpina M, Ahmed S, Ali AM, Mtoro AT, Hamad AS, Mutani P, Tanner M, Tinto H, D'Alessandro U, Sorgho H, Valea I, Bihoun B, Guiraud I, Kabore B, Sombie O, Guiguemde RT, Ouedraogo JB, Hamel MJ, Kariuki S, Oneko M, Odero C, Otieno K, Awino N, McMorrow M, Muturi-Kioi V, Laserson KF, Slutsker L, Otieno W, Otieno L, Otsyula N, Gondi S, Otieno A, Owira V, Oguk E, Odongo G, Woods JB, Ogutu B, Njuguna P, Chilengi R, Akoo P, Kerubo C, Maingi C, Lang T, Olotu A, Bejon P, Marsh K, Mwambingu G, Owusu-Agyei S, Asante KP, Osei-Kwakye K, Boahen O, Dosoo D, Asante I, Adjei G, Kwara E, Chandramohan D, Greenwood B, Lusingu J, Gesase S, Malabeja A, Abdul O, Mahende C, Liheluka E, Malle L, Lemnge M, Theander TG, Drakeley C, Ansong D, Agbenyega T, Adjei S, Boateng HO, Rettig T, Bawa J, Sylverken J, Sambian D, Sarfo A, Agyekum A, Martinson F, Hoffman I, Mvalo T, Kamthunzi P, Nkomo R, Tembo T, Tegha G, Tsidya M, Kilembe J, Chawinga C, Ballou WR, Cohen J, Guerra Y, Jongert E, Lapierre D, Leach A, Lievens M, Ofori-Anyinam O, Olivier A, Vekemans J, Carter T, Kaslow D, Leboulleux D, Loucq C, Radford A, Savarese B, Schellenberg D, Sillman M, Vansadia P. A phase 3 trial of RTS,S/AS01 malaria vaccine in African infants. N Engl J Med. 2012 Dec 13;367(24):2284-95. doi: 10.1056/NEJMoa1208394. Epub 2012 Nov 9. PMID 23136909
- [Background] RTS,S Clinical Trials Partnership; Agnandji ST, Lell B, Soulanoudjingar SS, Fernandes JF, Abossolo BP, Conzelmann C, Methogo BG, Doucka Y, Flamen A, Mordmuller B, Issifou S, Kremsner PG, Sacarlal J, Aide P, Lanaspa M, Aponte JJ, Nhamuave A, Quelhas D, Bassat Q, Mandjate S, Macete E, Alonso P, Abdulla S, Salim N, Juma O, Shomari M, Shubis K, Machera F, Hamad AS, Minja R, Mtoro A, Sykes A, Ahmed S, Urassa AM, Ali AM, Mwangoka G, Tanner M, Tinto H, D'Alessandro U, Sorgho H, Valea I, Tahita MC, Kabore W, Ouedraogo S, Sandrine Y, Guiguemde RT, Ouedraogo JB, Hamel MJ, Kariuki S, Odero C, Oneko M, Otieno K, Awino N, Omoto J, Williamson J, Muturi-Kioi V, Laserson KF, Slutsker L, Otieno W, Otieno L, Nekoye O, Gondi S, Otieno A, Ogutu B, Wasuna R, Owira V, Jones D, Onyango AA, Njuguna P, Chilengi R, Akoo P, Kerubo C, Gitaka J, Maingi C, Lang T, Olotu A, Tsofa B, Bejon P, Peshu N, Marsh K, Owusu-Agyei S, Asante KP, Osei-Kwakye K, Boahen O, Ayamba S, Kayan K, Owusu-Ofori R, Dosoo D, Asante I, Adjei G, Adjei G, Chandramohan D, Greenwood B, Lusingu J, Gesase S, Malabeja A, Abdul O, Kilavo H, Mahende C, Liheluka E, Lemnge M, Theander T, Drakeley C, Ansong D, Agbenyega T, Adjei S, Boateng HO, Rettig T, Bawa J, Sylverken J, Sambian D, Agyekum A, Owusu L, Martinson F, Hoffman I, Mvalo T, Kamthunzi P, Nkomo R, Msika A, Jumbe A, Chome N, Nyakuipa D, Chintedza J, Ballou WR, Bruls M, Cohen J, Guerra Y, Jongert E, Lapierre D, Leach A, Lievens M, Ofori-Anyinam O, Vekemans J, Carter T, Leboulleux D, Loucq C, Radford A, Savarese B, Schellenberg D, Sillman M, Vansadia P. First results of phase 3 trial of RTS,S/AS01 malaria vaccine in African children. N Engl J Med. 2011 Nov 17;365(20):1863-75. doi: 10.1056/NEJMoa1102287. Epub 2011 Oct 18. PMID 22007715
- [Background] Leach A, Vekemans J, Lievens M, Ofori-Anyinam O, Cahill C, Owusu-Agyei S, Abdulla S, Macete E, Njuguna P, Savarese B, Loucq C, Ballou WR; Clinical Trials Partnership Committee. Design of a phase III multicenter trial to evaluate the efficacy of the RTS,S/AS01 malaria vaccine in children across diverse transmission settings in Africa. Malar J. 2011 Aug 4;10:224. doi: 10.1186/1475-2875-10-224. PMID 21816029
- [Background] Lievens M, Aponte JJ, Williamson J, Mmbando B, Mohamed A, Bejon P, Leach A. Statistical methodology for the evaluation of vaccine efficacy in a phase III multi-centre trial of the RTS, S/AS01 malaria vaccine in African children. Malar J. 2011 Aug 4;10:222. doi: 10.1186/1475-2875-10-222. PMID 21816030
- [Background] Neafsey DE, Juraska M, Bedford T, Benkeser D, Valim C, Griggs A, Lievens M, Abdulla S, Adjei S, Agbenyega T, Agnandji ST, Aide P, Anderson S, Ansong D, Aponte JJ, Asante KP, Bejon P, Birkett AJ, Bruls M, Connolly KM, D'Alessandro U, Dobano C, Gesase S, Greenwood B, Grimsby J, Tinto H, Hamel MJ, Hoffman I, Kamthunzi P, Kariuki S, Kremsner PG, Leach A, Lell B, Lennon NJ, Lusingu J, Marsh K, Martinson F, Molel JT, Moss EL, Njuguna P, Ockenhouse CF, Ogutu BR, Otieno W, Otieno L, Otieno K, Owusu-Agyei S, Park DJ, Pelle K, Robbins D, Russ C, Ryan EM, Sacarlal J, Sogoloff B, Sorgho H, Tanner M, Theander T, Valea I, Volkman SK, Yu Q, Lapierre D, Birren BW, Gilbert PB, Wirth DF. Genetic Diversity and Protective Efficacy of the RTS,S/AS01 Malaria Vaccine. N Engl J Med. 2015 Nov 19;373(21):2025-2037. doi: 10.1056/NEJMoa1505819. Epub 2015 Oct 21. PMID 26488565
- [Background] RTS,S Clinical Trials Partnership. Efficacy and safety of the RTS,S/AS01 malaria vaccine during 18 months after vaccination: a phase 3 randomized, controlled trial in children and young infants at 11 African sites. PLoS Med. 2014 Jul 29;11(7):e1001685. doi: 10.1371/journal.pmed.1001685. eCollection 2014 Jul. PMID 25072396
- [Background] RTS,S Clinical Trials Partnership. Efficacy and safety of RTS,S/AS01 malaria vaccine with or without a booster dose in infants and children in Africa: final results of a phase 3, individually randomised, controlled trial. Lancet. 2015 Jul 4;386(9988):31-45. doi: 10.1016/S0140-6736(15)60721-8. Epub 2015 Apr 23. PMID 25913272
- [Background] Swysen C, Vekemans J, Bruls M, Oyakhirome S, Drakeley C, Kremsner P, Greenwood B, Ofori-Anyinam O, Okech B, Villafana T, Carter T, Savarese B, Duse A, Reijman A, Ingram C, Frean J, Ogutu B; Clinical Trials Partnership Committee. Development of standardized laboratory methods and quality processes for a phase III study of the RTS, S/AS01 candidate malaria vaccine. Malar J. 2011 Aug 4;10:223. doi: 10.1186/1475-2875-10-223. PMID 21816032
- [Background] Vandoolaeghe P, Schuerman L. The RTS,S/AS01 malaria vaccine in children 5 to 17 months of age at first vaccination. Expert Rev Vaccines. 2016 Dec;15(12):1481-1493. doi: 10.1080/14760584.2016.1236689. PMID 27841689
- [Background] Vekemans J, Marsh K, Greenwood B, Leach A, Kabore W, Soulanoudjingar S, Asante KP, Ansong D, Evans J, Sacarlal J, Bejon P, Kamthunzi P, Salim N, Njuguna P, Hamel MJ, Otieno W, Gesase S, Schellenberg D; Clinical Trials Partnership Committee. Assessment of severe malaria in a multicenter, phase III, RTS, S/AS01 malaria candidate vaccine trial: case definition, standardization of data collection and patient care. Malar J. 2011 Aug 4;10:221. doi: 10.1186/1475-2875-10-221. PMID 21816031
- [Derived] Potter GE, Callier V, Shrestha B, Joshi S, Dwivedi A, Silva JC, Laurens MB, Follmann DA, Deye GA. Can incorporating genotyping data into efficacy estimators improve efficiency of early phase malaria vaccine trials? Malar J. 2023 Dec 19;22(1):383. doi: 10.1186/s12936-023-04802-0. PMID 38115002
- [Derived] Potter GE, Callier V, Shrestha B, Joshi S, Dwivedi A, Silva JC, Laurens MB, Follmann DA, Deye GA. Can incorporating genotyping data into efficacy estimators improve efficiency of early phase malaria vaccine trials? Res Sq [Preprint]. 2023 Sep 22:rs.3.rs-3370731. doi: 10.21203/rs.3.rs-3370731/v1. PMID 37790581
- [Derived] Mwamlima TG, Mwakasungula SM, Mkindi CG, Tambwe MM, Mswata SS, Mbwambo SG, Mboya MF, Draper SJ, Silk SE, Mpina MG, Vianney JM, Olotu AI. Understanding the role of serological and clinical data on assessing the dynamic of malaria transmission: a case study of Bagamoyo district, Tanzania. Pan Afr Med J. 2022 Oct 7;43:60. doi: 10.11604/pamj.2022.43.60.35779. eCollection 2022. PMID 36578806
- [Derived] Moncunill G, Carnes J, Chad Young W, Carpp L, De Rosa S, Campo JJ, Nhabomba A, Mpina M, Jairoce C, Finak G, Haas P, Muriel C, Van P, Sanz H, Dutta S, Mordmuller B, Agnandji ST, Diez-Padrisa N, Williams NA, Aponte JJ, Valim C, Neafsey DE, Daubenberger C, McElrath MJ, Dobano C, Stuart K, Gottardo R. Transcriptional correlates of malaria in RTS,S/AS01-vaccinated African children: a matched case-control study. Elife. 2022 Jan 21;11:e70393. doi: 10.7554/eLife.70393. PMID 35060479
- [Derived] Gyaase S, Asante KP, Adeniji E, Boahen O, Cairns M, Owusu-Agyei S. Potential effect modification of RTS,S/AS01 malaria vaccine efficacy by household socio-economic status. BMC Public Health. 2021 Jan 28;21(1):240. doi: 10.1186/s12889-021-10294-x. PMID 33509156
- [Derived] Bell GJ, Loop MS, Mvalo T, Juliano JJ, Mofolo I, Kamthunzi P, Tegha G, Lievens M, Bailey J, Emch M, Hoffman I. Environmental modifiers of RTS,S/AS01 malaria vaccine efficacy in Lilongwe, Malawi. BMC Public Health. 2020 Jun 12;20(1):910. doi: 10.1186/s12889-020-09039-z. PMID 32532234
- [Derived] Otieno L, Guerra Mendoza Y, Adjei S, Agbenyega T, Agnandji ST, Aide P, Akoo P, Ansong D, Asante KP, Berkley JA, Gesase S, Hamel MJ, Hoffman I, Kaali S, Kamthunzi P, Kariuki S, Kremsner P, Lanaspa M, Lell B, Lievens M, Lusingu J, Malabeja A, Masoud NS, Mtoro AT, Njuguna P, Ofori-Anyinam O, Otieno GA, Otieno W, Owusu-Agyei S, Schuerman L, Sorgho H, Tanner M, Tinto H, Valea I, Vandoolaeghe P, Sacarlal J, Oneko M. Safety and immunogenicity of the RTS,S/AS01 malaria vaccine in infants and children identified as HIV-infected during a randomized trial in sub-Saharan Africa. Vaccine. 2020 Jan 22;38(4):897-906. doi: 10.1016/j.vaccine.2019.10.077. Epub 2019 Nov 7. PMID 31708182
- [Derived] Ward CL, Shaw D, Anane-Sarpong E, Sankoh O, Tanner M, Elger B. The Ethics of End-of-Trial Obligations in a Pediatric Malaria Vaccine Trial: The Perspectives of Stakeholders From Ghana and Tanzania. J Empir Res Hum Res Ethics. 2018 Jul;13(3):258-269. doi: 10.1177/1556264618771809. Epub 2018 May 13. PMID 29756531
- [Derived] Ward CL, Shaw D, Anane-Sarpong E, Sankoh O, Tanner M, Elger B. The Ethics of Health Care Delivery in a Pediatric Malaria Vaccine Trial: The Perspectives of Stakeholders From Ghana and Tanzania. J Empir Res Hum Res Ethics. 2018 Feb;13(1):26-41. doi: 10.1177/1556264617742236. Epub 2017 Nov 28. PMID 29179625
- [Derived] Ward CL, Shaw D, Anane-Sarpong E, Sankoh O, Tanner M, Elger B. Defining Health Research for Development: The perspective of stakeholders from an international health research partnership in Ghana and Tanzania. Dev World Bioeth. 2018 Dec;18(4):331-340. doi: 10.1111/dewb.12144. Epub 2017 May 3. PMID 28470856
- [Derived] Sauboin CJ, Van Bellinghen LA, Van De Velde N, Van Vlaenderen I. Potential public health impact of RTS,S malaria candidate vaccine in sub-Saharan Africa: a modelling study. Malar J. 2015 Dec 23;14:524. doi: 10.1186/s12936-015-1046-z. PMID 26702637
- [Derived] Angwenyi V, Kamuya D, Mwachiro D, Kalama B, Marsh V, Njuguna P, Molyneux S. Complex realities: community engagement for a paediatric randomized controlled malaria vaccine trial in Kilifi, Kenya. Trials. 2014 Feb 25;15:65. doi: 10.1186/1745-6215-15-65. PMID 24565019
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: 110021 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 110021 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 110021 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 110021 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 110021 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 110021 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study included 3 phases, a primary (PRI) phase (Months 0-3) and a booster (BST) phase at Month 20, each followed by a related PRI/BST efficacy, immunogenicity and safety (EIS) follow-up (FU) phase, and an EIS extension, from Month 32 to the median of Month 48 or Month 38 time point.
Pre-assignment Details: Screening included the following: check for inclusion/exclusion criteria, vaccination contraindications/precautions, subjects' medical history and signing informed consent forms.
Groups:
- GSK257049 [5-17M] Group: Male or female children between and including 5 to 17 months of age [5-17M], who received a 3-dose primary vaccination course of the GSK257049 malaria vaccine, according to a 0-1-2 Month schedule, followed by either a booster dose of the same GSK257049 vaccine or a dose of Menjugate® vaccine, at Month 20. Both vaccines have been administered intramuscularly into the left deltoid.
- GSK257049 [6-12W] Group: Male or female children between and including 6 to 12 weeks of age [6-12W], who received a 3-dose primary vaccination course of the GSK257049 malaria vaccine co-administered with Polio Sabin™ and Tritanrix HepB™/Hib vaccines, according to a 0-1-2 Month schedule, followed by either a booster dose of the GSK257049 and Polio Sabin™ vaccines or a booster dose of Menjugate® and Polio Sabin™ vaccines, at Month 20. All vaccines have been administered intramuscularly in the anterolateral left thigh (GSK257049 vaccine); left deltoid (GSK257049 booster dose); left thigh for children under 1 year and left deltoid for children above 1 year of age (Menjugate® vaccine); anterolateral right thigh (Tritanrix HepB™/Hib vaccine), except for the Polio Sabin™ vaccine, which has been given orally.
- VeroRab Comparator [5-17M] Group: Male or female children between and including 5 to 17 months of age [5-17M], who received a 3-dose primary vaccination course of the VeroRab® vaccine, according to a 0-1-2 Month schedule, followed by a booster dose of Menjugate® vaccine, at Month 20. Both vaccines have been administered intramuscularly into the left deltoid.
- Menjugate Comparator [6-12W] Group: Male or female children between and including 6 to 12 weeks of age [6-12W], who received a 3-dose primary vaccination course of Menjugate® vaccine co-administered with Polio Sabin™ and Tritanrix HepB™/Hib vaccines, according to a 0-1-2 Month schedule, followed by a booster dose of Menjugate® and Polio Sabin™ vaccines, at Month 12. All vaccines have been administered intramuscularly in the left thigh for children under 1 year and left deltoid for children above 1 year of age (Menjugate® vaccine); anterolateral right thigh (Tritanrix HepB™/Hib vaccine), except for the Polio Sabin™ vaccine, which has been given orally.
Period: Overall Study
Arm/Group | GSK257049 [5-17M] Group | GSK257049 [6-12W] Group | VeroRab Comparator [5-17M] Group | Menjugate Comparator [6-12W] Group
Started | 5948 | 4358 | 2974 | 2179
Completed | 4102 | 3088 | 2085 | 1549
Not Completed | 1846 | 1270 | 889 | 630
Not completed — Adverse Event | 112 | 106 | 47 | 44
Not completed — Protocol Violation | 2 | 39 | 2 | 17
Not completed — Withdrawal by Subject | 587 | 295 | 272 | 144
Not completed — Lost to Follow-up | 1145 | 830 | 568 | 425

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GSK257049 [5-17M] Group | GSK257049 [6-12W] Group | VeroRab Comparator [5-17M] Group | Menjugate Comparator [6-12W] Group | Total
Number analyzed (Participants) | 5948 | 4358 | 2974 | 2179 | 15459
Age, Continuous [Mean (Standard Deviation); unit: Months] | 10.6 (3.8) | 1.2 (0.4) | 10.6 (3.7) | 1.2 (0.4) | 6.6 (5.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2967 | 2124 | 1503 | 1100 | 7694
  Male | 2981 | 2234 | 1471 | 1079 | 7765
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African heritage/African American | 5948 | 4358 | 2974 | 2179 | 15459

OUTCOME MEASURES:

1. Primary Outcome: Rate of First or Only Clinical Episode of Plasmodium Falciparum (P. Falciparum) Malaria Infection (CPFMI), or Clinical Malaria Episode of Primary Case Definition (CPFMI-PCD)
Description: A CPFMI-PCD was defined as an episode of malaria for which P. falciparum asexual parasitemia was greater than (>) 5000 parasites per microliter (µL) accompanied by the presence of fever [axillary temperature greater than or equal to (≥) 37.5°C] at the time of presentation AND occurring in a child who is unwell and brought for treatment to a healthcare facility OR a case of malaria meeting the primary case definition of severe malaria disease. The time to first or only CPFMI-PCD is expressed in terms of rate of first or only CPFMI (RfoCPFMI), that is person-year rate in each group (n/T). Analysis for this outcome was solely performed on subjects in the 5-17 months age category.
Time Frame: From Month 2.5 to Month 14
Population: The analysis was performed on the According-to-Protocol (ATP) population for efficacy, which included all children aged 5-17 Months who received all vaccinations according to protocol procedures and contributed to the time at risk in the follow-up period starting 14 days post Dose 3.
Measure: Number; unit: events per person-year
Arm/Group | GSK257049 [5-17M] Group | VeroRab Comparator [5-17M] Group
Number analyzed (Participants) | 2830 | 1466
events per person-year | 0.435 | 0.833
Statistical Analysis 1: Comparison: GSK257049 [5-17M] Group vs VeroRab Comparator [5-17M] Group; The analysis aimed to compare RfoCPFMI between groups over the Months 2.5-14 time period. Using RfoCFPMI, a Cox regression model was used to evaluate vaccine efficacy (VE) allowing for adjustment by factors. VE was calculated as 1 minus [Hazard Ratio (HR) in GSK257049 [5-17M] Group (HR1) divided by HR in control VeroRab Comparator [5-17M] Group (HR2)]; i. e. 1 - (HR1/HR2); Test type: Superiority — Criterion for success = lower limit (LL) of 97.5% confidence interval (CI) of VE > 0; p < 0.0001, Regression, Cox; Vaccine efficacy = 55.8, 97.5% CI 2-sided [50.6 to 60.4]

2. Primary Outcome: Rate of First or Only Clinical Episode of P. Falciparum Malaria Infection (CPFMI), or Clinical Malaria Episode of Primary Case Definition (CPFMI-PCD)
Description: A CPFMI-PCD was defined as an episode of malaria for which P. falciparum asexual parasitemia > 5000 parasites/µL was accompanied by the presence of fever (axillary temperature ≥ 37.5°C) at the time of presentation AND occurring in a child who is unwell and brought for treatment to a healthcare facility OR a case of malaria meeting the primary case definition of severe malaria disease. The time to first or only CPFMI-PCD is expressed in terms of rate of first or only CPFMI (RfoCPFMI), that is, person-year rate in each group (n/T). Analysis for this outcome was solely performed on subjects in the 6-12 weeks (6-12W) age category.
Time Frame: From Month 2.5 to Month 14
Population: The analysis was performed on the ATP population for efficacy, which included all children aged 6-12 Weeks who received all vaccinations according to protocol procedures and contributed to the time at risk in the follow-up period starting 14 days post Dose 3.
Measure: Number; unit: events per person-year
Arm/Group | GSK257049 [6-12W] Group | Menjugate Comparator [6-12W] Group
Number analyzed (Participants) | 3995 | 2008
events per person-year | 0.367 | 0.484
Statistical Analysis 1: Comparison: GSK257049 [6-12W] Group vs Menjugate Comparator [6-12W] Group; The analysis aimed to compare RfoCPFMI between groups over the Months 2.5-14 time period. Using RfoCFPMI, a Cox regression model was used to evaluate vaccine efficacy (VE) allowing for adjustment by factors. VE was calculated as 1 minus [Hazard Ratio (HR) in GSK257049 [6-12W] Group (HR1) divided by HR in control Menjugate Comparator [6-12W] Group (HR2)]; i. e. 1 - (HR1/HR2); Test type: Superiority — Point estimate of efficacy was adjusted for study site as stratification factor for the analysis. Criterion for success = lower limit (LL) of 97.5% confidence interval (CI) of VE > 0; p < 0.0001, Regression, Cox; Vaccine efficacy = 31.315, 97.5% CI 2-sided [23.556 to 38.286]

3. Secondary Outcome: Rate of All Episodes of P. Falciparum Clinical Malaria Infection (CPFMI) of PCD and of Secondary Case Definitions (SCD) 1, SCD 2 and SCD 3
Description: PCD=malaria episode with P. falciparum asexual parasitemia (PFAP) > 5000 parasites/µL accompanied by fever and occurring in a child unwell brought for treatment to a healthcare facility or a case of malaria meeting the PCD of severe malaria disease. SCD1=malaria episode with PFAP > 0 and fever at time of presentation or history of fever within 24h of presentation in a subject unwell brought for treatment to a healthcare facility. SCD2=malaria episode with PFAP > 500 parasites/μL and fever at time of presentation in a subject unwell brought for treatment to a healthcare facility. SCD3=malaria episode with PFAP > 20.000 parasites/μL and fever at time of presentation in a subject unwell and brought for treatment to a healthcare facility. Time to all CPFMI episodes is expressed as person-year rate in each group (n/T). Results are uncorrected for double enrollment of 1 subject receiving GSK257049 vaccine.
Time Frame: From Month 2.5 to Month 14
Population: The analysis was performed on the ATP population for efficacy, which included all children who received all vaccinations according to protocol procedures and contributed to the time at risk in the follow-up period starting 14 days post Dose 3.
Measure: Number; unit: events per person-year
Arm/Group | GSK257049 [5-17M] Group | GSK257049 [6-12W] Group | VeroRab Comparator [5-17M] Group | Menjugate Comparator [6-12W] Group
Number analyzed (Participants) | 2830 | 3995 | 1466 | 2008
events per person-year
  PCD | 0.735 | 0.639 | 1.468 | 0.908
  SCD1 | 1.224 | 0.989 | 2.312 | 1.403
  SCD2 | 0.847 | 0.736 | 1.628 | 1.031
  SCD3 | 0.625 | 0.515 | 1.244 | 0.731

4. Secondary Outcome: Rate of All Episodes of Clinical P. Falciparum Malaria Infection (CPFMI) of PCD, Overall and by Center
Description: PCD = malaria episode with PFAP > 5000 parasites/µL accompanied by fever and occurring in a child unwell brought for treatment to a healthcare facility or a case of malaria meeting the PCD of severe malaria disease (see below endpoints on severe malaria for details). Time to all CPFMI episodes is expressed as person-year rate in each group (n/T). Results are by center and across centers, and are uncorrected for double enrollment of 1 subject receiving GSK257049 vaccine.
Time Frame: From Month 2.5 to Month 20
Population: The analysis was performed on the ATP population for efficacy, which included all children who received all vaccinations according to protocol procedures and contributed to the time at risk in the follow-up period starting 14 days post Dose 3. Data was not collected for the participants in the 5-17M groups for the Manhica site.
Measure: Number; unit: events per person-year
Arm/Group | GSK257049 [5-17M] Group | GSK257049 [6-12W] Group | VeroRab Comparator [5-17M] Group | Menjugate Comparator [6-12W] Group
Number analyzed (Participants) | 4557 | 3996 | 2328 | 2007
events per person-year
  PCD - Agogo: number analyzed (Participants) | 371 | 418 | 192 | 221
  PCD - Agogo | 0.56 | 0.64 | 1.16 | 0.79
  PCD - Bagamoyo: number analyzed (Participants) | 462 | 502 | 235 | 244
  PCD - Bagamoyo | 0.1 | 0.08 | 0.28 | 0.14
  PCD - Kilifi: number analyzed (Participants) | 336 | 186 | 171 | 102
  PCD - Kilifi | 0.01 | 0.04 | 0.04 | 0.02
  PCD - Kintampo: number analyzed (Participants) | 602 | 199 | 296 | 99
  PCD - Kintampo | 1.01 | 1.53 | 1.85 | 1.49
  PCD - Kombewa: number analyzed (Participants) | 609 | 387 | 311 | 196
  PCD - Kombewa | 1.21 | 0.94 | 1.87 | 1.32
  PCD - Korogwe: number analyzed (Participants) | 568 | 382 | 293 | 183
  PCD - Korogwe | 0.04 | 0.03 | 0.11 | 0.05
  PCD - Lambarene: number analyzed (Participants) | 380 | 147 | 196 | 62
  PCD - Lambarene | 0.11 | 0.11 | 0.2 | 0.12
  PCD - Lilongwe: number analyzed (Participants) | 359 | 500 | 183 | 258
  PCD - Lilongwe | 0.2 | 0.3 | 0.32 | 0.5
  PCD - Manhica: number analyzed (Participants) | 0 | 381 | 0 | 188
  PCD - Manhica |  | 0.1 |  | 0.12
  PCD - Nanoro: number analyzed (Participants) | 389 | 441 | 198 | 225
  PCD - Nanoro | 1.42 | 1.93 | 2.4 | 2.39
  PCD - Siaya: number analyzed (Participants) | 481 | 453 | 253 | 229
  PCD - Siaya | 2.01 | 2.03 | 3.31 | 2.75
  PCD - Across | 0.69 | 0.71 | 1.17 | 0.92

5. Secondary Outcome: Rate of All Episodes of Clinical P. Falciparum Malaria Infection (CPFMI) of SCD1, SCD2 and SCD3 (Overall)
Description: SCD1 = malaria episode with PFAP > 0 and fever at time of presentation or history of fever within 24h of presentation in a subject unwell brought for treatment to a healthcare facility. SCD2 = malaria episode with PFAP > 500 parasites/μL and fever at time of presentation in a subject unwell brought for treatment to a healthcare facility. SCD3 = malaria episode with PFAP > 20.000 parasites/μL and fever at time of presentation in a subject unwell and brought for treatment to a healthcare facility. Time to all CPFMI episodes is expressed as person-year rate in each group (n/T). Results are across centers, and are uncorrected for double enrollment of 1 subject receiving GSK257049 vaccine.
Time Frame: From Month 2.5 to Month 20
Population: as for outcome 3
Measure: Number; unit: events per person-year
Arm/Group | GSK257049 [5-17M] Group | GSK257049 [6-12W] Group | VeroRab Comparator [5-17M] Group | Menjugate Comparator [6-12W] Group
Number analyzed (Participants) | 4557 | 3996 | 2328 | 2007
events per person-year
  SCD1 | 1.09 | 1.09 | 1.78 | 1.42
  SCD2 | 0.78 | 0.81 | 1.3 | 1.04
  SCD3 | 0.59 | 0.58 | 1.01 | 0.76

6. Secondary Outcome: Rate of All Episodes of Clinical P. Falciparum Malaria Infection (CPFMI) of Primary Case Definition (PCD), by Centers and Across Centers
Description: CPFMI of PCD = episode of malaria for which PFAP > 5000 parasites/µL accompanied by presence of fever (axillary temperature ≥ 37.5°C at time of presentation) AND occurring in a child unwell brought for treatment to a healthcare facility OR a case of malaria meeting the PCD of severe malaria disease. Time to all CPFMI episodes is expressed as person-year rate in each group (n/T). Results are presented by center and across centers.
Time Frame: From Month 2.5 up to study End (with a median follow-up time post-Dose 1 of 48 months for 5-17M groups and 38 months for 6-12W groups)
Population: as for outcome 4
Measure: Number; unit: events per person-year
Groups:
- GSK257049 - GSK257049 [5-17M] Group: Male or female children between and including 5 to 17 months of age [5-17M], who received a 3-dose primary vaccination course of the GSK257049 malaria vaccine, according to a 0-1-2 Month schedule, followed by a booster dose of the same GSK257049 vaccine, at Month 20. Both vaccines have been administered intramuscularly into the left deltoid.
- GSK257049 - Menjugate [5-17M] Group: Male or female children between and including 5 to 17 months of age [5-17M], who received a 3-dose primary vaccination course of the GSK257049 malaria vaccine, according to a 0-1-2 Month schedule, followed by a booster dose of Menjugate® vaccine, at Month 20. Both vaccines have been administered intramuscularly into the left deltoid.
- GSK257049 -GSK257049 [6-12W] Group: Male or female children between and including 6 to 12 weeks of age [6-12W], who received a 3-dose primary vaccination course of the GSK257049 malaria vaccine co-administered with Polio Sabin™ and Tritanrix HepB™/Hib vaccines, according to a 0-1-2 Month schedule, followed by a booster dose of the GSK257049 and Polio Sabin™ vaccines, at Month 20. All vaccines have been administered intramuscularly in the anterolateral left thigh (GSK257049 vaccine); left deltoid (GSK257049 booster dose); anterolateral right thigh (Tritanrix HepB™/Hib vaccine), except for the Polio Sabin™ vaccine, which has been given orally.
- GSK257049 - Menjugate [6-12W] Group: Male or female children between and including 6 to 12 weeks of age [6-12W], who received a 3-dose primary vaccination course of the GSK257049 malaria vaccine co-administered with Polio Sabin™ and Tritanrix HepB™/Hib vaccines, according to a 0-1-2 Month schedule, followed by a booster dose of Menjugate® and Polio Sabin™ vaccines, at Month 20. All vaccines have been administered intramuscularly in the anterolateral left thigh (GSK257049 vaccine); left deltoid (GSK257049 booster dose); left thigh for children under 1 year and left deltoid for children above 1 year of age (Menjugate® vaccine); anterolateral right thigh (Tritanrix HepB™/Hib vaccine), except for the Polio Sabin™ vaccine, which has been given orally.
Arm/Group | GSK257049 - GSK257049 [5-17M] Group | GSK257049 - Menjugate [5-17M] Group | VeroRab Comparator [5-17M] Group | GSK257049 -GSK257049 [6-12W] Group | GSK257049 - Menjugate [6-12W] Group | Menjugate Comparator [6-12W] Group
Number analyzed (Participants) | 2276 | 2306 | 2336 | 1985 | 2005 | 2007
events per person-year
  PCD - Kilifi: number analyzed (Participants) | 163 | 172 | 172 | 90 | 95 | 102
  PCD - Kilifi | 0.02 | 0.03 | 0.08 | 0.06 | 0.04 | 0.04
  PCD - Korogwe: number analyzed (Participants) | 286 | 282 | 293 | 191 | 191 | 183
  PCD - Korogwe | 0.04 | 0.05 | 0.1 | 0.05 | 0.07 | 0.09
  PCD - Lambarene: number analyzed (Participants) | 187 | 196 | 196 | 72 | 75 | 62
  PCD - Lambarene | 0.15 | 0.15 | 0.23 | 0.1 | 0.18 | 0.17
  PCD - Bagamoyo: number analyzed (Participants) | 228 | 242 | 236 | 252 | 249 | 245
  PCD - Bagamoyo | 0.16 | 0.21 | 0.27 | 0.08 | 0.11 | 0.15
  PCD - Lilongwe: number analyzed (Participants) | 176 | 183 | 185 | 247 | 250 | 257
  PCD - Lilongwe | 0.09 | 0.2 | 0.23 | 0.25 | 0.29 | 0.42
  PCD - Agogo: number analyzed (Participants) | 188 | 183 | 191 | 209 | 209 | 221
  PCD - Agogo | 0.59 | 0.73 | 1.01 | 0.59 | 0.77 | 0.84
  PCD - Kombewa: number analyzed (Participants) | 315 | 301 | 312 | 195 | 193 | 196
  PCD - Kombewa | 1.26 | 1.37 | 1.64 | 1.37 | 1.37 | 1.62
  PCD - Kintampo: number analyzed (Participants) | 299 | 310 | 301 | 98 | 101 | 100
  PCD - Kintampo | 1.11 | 1.31 | 1.71 | 1.65 | 1.71 | 1.69
  PCD - Manhica: number analyzed (Participants) | 0 | 0 | 0 | 193 | 187 | 188
  PCD - Manhica |  |  |  | 0.18 | 0.14 | 0.2
  PCD - Nanoro: number analyzed (Participants) | 194 | 195 | 198 | 217 | 224 | 224
  PCD - Nanoro | 1.95 | 2.18 | 2.69 | 2.59 | 2.79 | 3.14
  PCD - Siaya: number analyzed (Participants) | 240 | 242 | 252 | 221 | 231 | 229
  PCD - Siaya | 2.09 | 2.55 | 3.15 | 2.43 | 2.67 | 3.12
  PCD - Across | 0.79 | 0.9 | 1.14 | 0.86 | 0.95 | 1.08

7. Secondary Outcome: Rate of All Episodes of Clinical P. Falciparum Malaria Infection (CPFMI) of Secondary Case Definition 1 (SCD1), Across Centers
Description: CPFMI of SCD1 = malaria episode with PFAP >0 and fever at time of presentation or history of fever within 24h of presentation in a subject unwell brought for treatment to a healthcare facility. Time to all CPFMI episodes is expressed as person-year rate in each group (n/T). Results are presented across centers.
Time Frame: as for outcome 6
Population: as for outcome 3
Measure: Number; unit: events per person-year
Arm/Group | GSK257049 - GSK257049 [5-17M] Group | GSK257049 - Menjugate [5-17M] Group | VeroRab Comparator [5-17M] Group | GSK257049 -GSK257049 [6-12W] Group | GSK257049 - Menjugate [6-12W] Group | Menjugate Comparator [6-12W] Group
Number analyzed (Participants) | 2276 | 2306 | 2336 | 1985 | 2005 | 2007
events per person-year | 1.26 | 1.41 | 1.81 | 1.29 | 1.43 | 1.61

8. Secondary Outcome: Rate of All Episodes of Clinical P. Falciparum Malaria Infection (CPFMI) of Primary Case Definition (PCD) and Secondary Case Definition 1 (SCD1), Across Centers
Description: CPFMI of PCD = episode of malaria for which PFAP > 5000 parasites/µL accompanied by the presence of fever (axillary temperature ≥ 37.5°C at time of presentation) AND occurring in a child unwell brought for treatment to a healthcare facility OR a case of malaria meeting the PCD of severe malaria disease. CPFMI of SCD1 = malaria episode with PFAP >0 and fever at time of presentation or history of fever within 24h of presentation in a subject unwell brought for treatment to a healthcare facility. Time to all CPFMI episodes is expressed as person-year rate in each group (n/T). Results are presented across centers.
Time Frame: From Booster at Month 20 up to study end (with a median follow-up time post-Dose 1 of 48 months for 5-17M groups and 38 months for 6-12W groups)
Population: as for outcome 3
Measure: Number; unit: events per person-year
Arm/Group | GSK257049 - GSK257049 [5-17M] Group | GSK257049 - Menjugate [5-17M] Group | VeroRab Comparator [5-17M] Group | GSK257049 -GSK257049 [6-12W] Group | GSK257049 - Menjugate [6-12W] Group | Menjugate Comparator [6-12W] Group
Number analyzed (Participants) | 2017 | 2057 | 2050 | 1743 | 1788 | 1762
events per person-year
  PCD | 0.87 | 1.03 | 1.1 | 1.01 | 1.21 | 1.23
  SCD1 | 1.39 | 1.65 | 1.82 | 1.48 | 1.79 | 1.8

9. Secondary Outcome: Rate of All Episodes of Clinical P. Falciparum Malaria Infection (CPFMI) of PCD and SCD1, Across Centers
Description: CPFMI of PCD = episode of malaria for which PFAP > 5000 parasites/µL accompanied by the presence of fever (axillary temperature ≥ 37.5°C at time of presentation) AND occurring in a child unwell brought for treatment to a healthcare facility OR a case of malaria meeting the PCD of severe malaria disease. CPFMI of SCD1 = malaria episode with PFAP > 0 and fever at time of presentation or history of fever within 24h of presentation in a subject unwell brought for treatment to a healthcare facility. Time to all CPFMI episodes is expressed as person-year rate in each group (n/T). Results are presented across centers.
Time Frame: From Month 33 up to study end (with a median follow-up time post-Dose 1 of 48 months for 5-17M groups and 38 months for 6-12W groups)
Population: as for outcome 3
Measure: Number; unit: events per person-year
Arm/Group | GSK257049 - GSK257049 [5-17M] Group | GSK257049 - Menjugate [5-17M] Group | VeroRab Comparator [5-17M] Group | GSK257049 -GSK257049 [6-12W] Group | GSK257049 - Menjugate [6-12W] Group | Menjugate Comparator [6-12W] Group
Number analyzed (Participants) | 1784 | 1838 | 1864 | 1516 | 1548 | 1546
events per person-year
  PCD | 1.01 | 1.1 | 1.1 | 1.18 | 1.31 | 1.29
  SCD1: number analyzed (Participants) | 1784 | 1838 | 1864 | 1516 | 1547 | 1546
  SCD1 | 1.61 | 1.79 | 1.88 | 1.73 | 1.92 | 1.91

10. Secondary Outcome: Rate of All Episodes of Clinical P. Falciparum Malaria Infection (CPFMI) of PCD, by Center and Across Centers
Description: CPFMI of PCD = episode of malaria for which PFAP > 5000 parasites/µL accompanied by the presence of fever (axillary temperature ≥ 37.5°C at time of presentation) AND occurring in a child unwell brought for treatment to a healthcare facility OR a case of malaria meeting the PCD of severe malaria disease. Time to all CPFMI episodes is expressed as person-year rate in each group (n/T). Results are presented by center and across centers.
Time Frame: From Month 2.5 to Month 32
Population: as for outcome 4
Measure: Number; unit: events per person-year
Arm/Group | GSK257049 - GSK257049 [5-17M] Group | GSK257049 - Menjugate [5-17M] Group | VeroRab Comparator [5-17M] Group | GSK257049 -GSK257049 [6-12W] Group | GSK257049 - Menjugate [6-12W] Group | Menjugate Comparator [6-12W] Group
Number analyzed (Participants) | 2276 | 2306 | 2336 | 1985 | 2005 | 2007
events per person-year
  PCD - Kilifi: number analyzed (Participants) | 163 | 172 | 172 | 90 | 95 | 102
  PCD - Kilifi | 0.03 | 0.04 | 0.09 | 0.06 | 0.04 | 0.05
  PCD - Korogwe: number analyzed (Participants) | 286 | 282 | 293 | 191 | 191 | 183
  PCD - Korogwe | 0.04 | 0.03 | 0.08 | 0.02 | 0.06 | 0.06
  PCD - Lambarene: number analyzed (Participants) | 187 | 196 | 196 | 72 | 75 | 62
  PCD - Lambarene | 0.14 | 0.14 | 0.21 | 0.1 | 0.18 | 0.18
  PCD - Bagamoyo: number analyzed (Participants) | 228 | 242 | 236 | 252 | 249 | 245
  PCD - Bagamoyo | 0.13 | 0.19 | 0.31 | 0.08 | 0.11 | 0.15
  PCD - Lilongwe: number analyzed (Participants) | 176 | 183 | 185 | 247 | 250 | 257
  PCD - Lilongwe | 0.11 | 0.22 | 0.29 | 0.27 | 0.32 | 0.47
  PCD - Agogo: number analyzed (Participants) | 188 | 183 | 191 | 209 | 209 | 221
  PCD - Agogo | 0.59 | 0.75 | 1.15 | 0.56 | 0.72 | 0.86
  PCD - Kombewa: number analyzed (Participants) | 315 | 301 | 312 | 195 | 193 | 196
  PCD - Kombewa | 1.12 | 1.29 | 1.67 | 1.28 | 1.25 | 1.55
  PCD - Kintampo: number analyzed (Participants) | 299 | 310 | 301 | 98 | 101 | 100
  PCD - Kintampo | 1.08 | 1.17 | 1.87 | 1.52 | 1.6 | 1.6
  PCD - Manhica: number analyzed (Participants) | 0 | 0 | 0 | 193 | 187 | 188
  PCD - Manhica |  |  |  | 0.15 | 0.12 | 0.15
  PCD - Nanoro: number analyzed (Participants) | 194 | 195 | 198 | 217 | 224 | 224
  PCD - Nanoro | 1.42 | 1.67 | 2.45 | 2.27 | 2.53 | 2.92
  PCD - Siaya: number analyzed (Participants) | 240 | 242 | 252 | 221 | 231 | 229
  PCD - Siaya | 1.91 | 2.46 | 3.25 | 2.41 | 2.54 | 3.09
  PCD - Across | 0.68 | 0.81 | 1.15 | 0.8 | 0.88 | 1.03

11. Secondary Outcome: Rate of All Episodes of Clinical P. Falciparum Malaria Infection (CPFMI) of Secondary Case Definition 1 (SCD1)
Description: CPFMI of SCD1 = malaria episode with PFAP > 0 and fever at time of presentation or history of fever within 24h of presentation in a subject unwell brought for treatment to a healthcare facility. Time to all episodes of CPFMI is expressed as a rate of all CPFMI (RaCPFMI), that is, person-year rate in each group (n/T).
Time Frame: From Month 2.5 to Month 32
Population: as for outcome 3
Measure: Number; unit: events per person-year
Arm/Group | GSK257049 - GSK257049 [5-17M] Group | GSK257049 - Menjugate [5-17M] Group | VeroRab Comparator [5-17M] Group | GSK257049 -GSK257049 [6-12W] Group | GSK257049 - Menjugate [6-12W] Group | Menjugate Comparator [6-12W] Group
Number analyzed (Participants) | 2276 | 2306 | 2336 | 1985 | 2005 | 2007
events per person-year | 1.1 | 1.24 | 1.78 | 1.19 | 1.33 | 1.54

12. Secondary Outcome: Rate of All Episodes of Clinical P. Falciparum Malaria Infection (CPFMI) of Primary Case Definition (PCD) and Secondary Case Definition 1 (SCD1)
Description: CPFMI of PCD = episode of malaria for which PFAP > 5000 parasites/µL accompanied by the presence of fever (axillary temperature ≥ 37.5°C at time of presentation) AND occurring in a child unwell brought for treatment to a healthcare facility OR a case of malaria meeting the PCD of severe malaria disease. CPFMI of SCD1 = malaria episode with PFAP > 0 and fever at time of presentation or history of fever within 24h of presentation in a subject unwell brought for treatment to a healthcare facility. Time to all episodes of CPFMI is expressed as a rate of all CPFMI (RaCPFMI), that is, person-year rate in each group (n/T).
Time Frame: From Booster at Month 20 up to Month 32
Population: as for outcome 3
Measure: Number; unit: events per person-year
Arm/Group | GSK257049 - GSK257049 [5-17M] Group | GSK257049 - Menjugate [5-17M] Group | VeroRab Comparator [5-17M] Group | GSK257049 -GSK257049 [6-12W] Group | GSK257049 - Menjugate [6-12W] Group | Menjugate Comparator [6-12W] Group
Number analyzed (Participants) | 2017 | 2057 | 2050 | 1743 | 1788 | 1762
events per person-year
  PCD | 0.72 | 0.96 | 1.1 | 0.91 | 1.15 | 1.2
  SCD1 | 1.14 | 1.48 | 1.74 | 1.35 | 1.72 | 1.74

13. Secondary Outcome: Percentage of Subjects With Severe PFMI (SPFMI) of PCD, SCD1, SCD2 and SCD3, Across Centers
Description: SPFMI of PCD = PFMI > 5000 parasites/μL, at least one severity marker and no co-morbidity diagnosis. SPFMI of SCD1 = PFMI >5000 parasites/μL and with one or more severity marker. SPFMI of SCD2 = PFMI >0 with one or more severity marker and without co-morbidity diagnosis. SPFMI of SCD3 = PFMI >5000 parasites/μL, with one or more severity marker, and without co-morbidity or HIV. Severity markers = prostration; respiratory distress; Blantyre score ≤ 2; ≥ 2 seizures in 24 h prior to admission, emergency room and hospitalisation; hypoglycaemia < 2.2 mmol/L; acidosis BE ≤ -10.0 mmol/L,l < 5.0 mmol/L; anaemia<5.0 g/dL. Comorbidities = radiographically proven pneumonia; meningitis; positive blood culture on a blood culture taken within 72 h of admission; gastroenteritis with dehydration. Analysis was performed in a pooled manner across age categories. Results presented are uncorrected for double enrollment of one subject in 5-17 months age category receiving GSK257049 vaccine.
Time Frame: From Month 2.5 up to the time when 250 subjects were diagnosed with severe malaria of PCD, SCD1, SCD2 and SCD3 (up to the Month 14 time point for each age category or date of booster dose, whichever occurred first)
Population: The analysis was performed, across age categories for which groups were pooled from the ATP population for efficacy. This included all children who received all vaccinations according to protocol procedures and contributed to the time at risk in the follow-up period starting 14 days post Dose 3.
Measure: Number; unit: Percentage of subjects
Groups:
- GSK257049 Group: For the purpose of the analysis, GSK257049 [5-17M] and GSK257049 [6-12W] groups have been pooled into a single group.
- Comparator Group: For the purpose of the analysis, VeroRab Comparator [5-17M] and Menjugate Comparator [6-12W] groups have been pooled into a single group.
Arm/Group | GSK257049 Group | Comparator Group
Number analyzed (Participants) | 8597 | 4364
Percentage of subjects
  PCD | 0.019 | 0.03
  SCD1 | 0.023 | 0.036
  SCD2 | 0.023 | 0.034
  SCD3 | 0.019 | 0.03

14. Secondary Outcome: Percentage of Subjects With Severe PFMI (SPFMI) of PCD and SCD1
Description: SPFMI of PCD = PFMI>5000 parasites/μL, at least one severity marker and no co-morbidity diagnosis. SPFMI of SCD1 = PFMI>5000 parasites/μL and with one or more severity marker. Severity markers = prostration; respiratory distress; Blantyre score ≤ 2; ≥ 2 seizures in 24h prior to admission, emergency room and hospitalisation; hypoglycaemia<2.2 mmol/L; acidosis BE ≤ -10.0 mmol/L,l ≥ 5.0 mmol/L; anaemia<5.0 g/dL. Comorbidities = radiographically proven pneumonia; meningitis; positive blood culture on a blood culture taken within 72h of admission; gastroenteritis with dehydration. SPFMI of SCD1 = PFMI>5000 parasites/μL and with one or more severity marker. Severity markers = prostration; respiratory distress; Blantyre score ≤ 2; ≥ 2 seizures in 24h prior to admission, emergency room and hospitalisation; hypoglycaemia<2.2 mmol/L; acidosis BE ≤ -10.0 mmol/L,l ≥ 5.0 mmol/L; anaemia<5.0 g/dL. Results presented are uncorrected for double enrollment of one subject in 5-17 months age category.
Time Frame: From Month 2.5 to Month 14
Population: as for outcome 3
Measure: Number; unit: Percentage of subjects
Arm/Group | GSK257049 [5-17M] Group | GSK257049 [6-12W] Group | VeroRab Comparator [5-17M] Group | Menjugate Comparator [6-12W] Group
Number analyzed (Participants) | 2830 | 3995 | 1466 | 2008
Percentage of subjects
  SPFMI PCD | 2.0 | 1.5 | 3.8 | 2.3
  SPFMI SCD1 | 2.6 | 1.6 | 4.9 | 2.5

15. Secondary Outcome: Percentage of Subjects With Severe PFMI (SPFMI) of PCD and SCD1
Description: as for outcome 14
Time Frame: From Month 2.5 to Month 20 at Booster
Population: as for outcome 3
Measure: Number; unit: Percentage of subjects
Arm/Group | GSK257049 [5-17M] Group | GSK257049 [6-12W] Group | VeroRab Comparator [5-17M] Group | Menjugate Comparator [6-12W] Group
Number analyzed (Participants) | 4557 | 3996 | 2328 | 2007
Percentage of subjects
  SPFMI PCD | 0.03 | 0.03 | 0.04 | 0.03
  SPFMI SCD1 | 0.03 | 0.03 | 0.05 | 0.03

16. Secondary Outcome: Percentage of Subjects With Severe PFMI (SPFMI) of PCD and SCD1
Description: SPFMI of PCD = PFMI >5000 parasites/μL, at least one severity marker and no co-morbidity diagnosis. SPFMI of SCD1 = PFMI >5000 parasites/μL and with one or more severity marker. Severity markers = prostration; respiratory distress; Blantyre score ≤ 2; ≥ 2 seizures in 24 h prior to admission, emergency room and hospitalisation; hypoglycaemia<2.2 mmol/L; acidosis BE ≤ -10.0 mmol/L,l ≥ 5.0 mmol/L; anaemia<5.0 g/dL. Comorbidities = radiographically proven pneumonia; meningitis; positive blood culture on a blood culture taken within 72 h of admission; gastroenteritis with dehydration. SPFMI of SCD1 = PFMI >5000 parasites/μL and with one or more severity marker. Severity markers = prostration; respiratory distress; Blantyre score ≤ 2; ≥ 2 seizures in 24 h prior to admission, emergency room and hospitalisation; hypoglycaemia<2.2 mmol/L; acidosis BE ≤ -10.0 mmol/L,l ≥ 5.0 mmol/L; anaemia<5.0 g/dL.
Time Frame: From Month 2.5, from Month 20(booster), from Month 33 up to study end (median follow-up time of 48 months post-Dose 1 for 5-17M age category and of 38 months post-Dose 1 for 6-12W age category) and from Month 2.5 to Month 32 and from Month 20 to Month 32
Population: as for outcome 3
Measure: Number; unit: Percentage of subjects
Arm/Group | GSK257049 - GSK257049 [5-17M] Group | GSK257049 - Menjugate [5-17M] Group | VeroRab Comparator [5-17M] Group | GSK257049 -GSK257049 [6-12W] Group | GSK257049 - Menjugate [6-12W] Group | Menjugate Comparator [6-12W] Group
Number analyzed (Participants) | 2276 | 2306 | 2336 | 1985 | 2005 | 2007
Percentage of subjects
  PCD, M2.5 to SE | 0.04 | 0.06 | 0.06 | 0.04 | 0.04 | 0.05
  PCD, M20 to SE: number analyzed (Participants) | 2017 | 2057 | 2051 | 1743 | 1788 | 1762
  PCD, M20 to SE | 0.03 | 0.04 | 0.02 | 0.02 | 0.03 | 0.03
  PCD, M33 to SE: number analyzed (Participants) | 1784 | 1838 | 1864 | 1516 | 1548 | 1546
  PCD, M33 to SE | 0.01 | 0.02 | 0.01 | 0.01 | 0.01 | 0.01
  PCD, M2.5 to M32 | 0.03 | 0.05 | 0.05 | 0.04 | 0.04 | 0.04
  PCD, M20 to M32: number analyzed (Participants) | 2017 | 2057 | 2051 | 1743 | 1788 | 1762
  PCD, M20 to M32 | 0.02 | 0.02 | 0.02 | 0.01 | 0.02 | 0.02
  SCD1, M2.5 to SE | 0.05 | 0.07 | 0.07 | 0.04 | 0.05 | 0.06
  SCD1, M20 to SE: number analyzed (Participants) | 2017 | 2057 | 2051 | 1743 | 1788 | 1762
  SCD1, M20 to SE | 0.03 | 0.04 | 0.03 | 0.02 | 0.03 | 0.03
  SCD1, M33 to SE: number analyzed (Participants) | 1784 | 1838 | 1864 | 1516 | 1548 | 1546
  SCD1, M33 to SE | 0.01 | 0.02 | 0.01 | 0.01 | 0.01 | 0.01
  SCD1, M2.5 to M32 | 0.04 | 0.06 | 0.06 | 0.04 | 0.04 | 0.05
  SCD1, M20 to M32: number analyzed (Participants) | 2017 | 2057 | 2051 | 1743 | 1788 | 1762
  SCD1, M20 to M32 | 0.02 | 0.03 | 0.02 | 0.01 | 0.02 | 0.02

17. Secondary Outcome: Percentage of Subjects With Incident Severe Anaemia (ISA) and Malaria Hospitalization (MH) for Case Definitions (CD) Considered
Description: CD considered were CD1 for ISA and CD1 and CD2 for MH. ISA of CD1 was defined as a documented hemoglobin < 5.0 g/dL identified at clinical presentation to morbidity surveillance system in association with a P. falciparum parasitemia > 5000 parasites/μL. MH of CD1 was defined as a medical hospitalization with confirmed P. falciparum > 5000 parasites/μL. MH of CD2 was defined as a hospitalization which, in the judgment of the principal investigator, P. falciparum infection was the sole or a major contributing factor to the presentation. Results presented are uncorrected for double enrollment of one subject in 5-17 months age category receiving GSK257049 vaccine.
Time Frame: From Month 2.5 to Month 20
Population: as for outcome 3
Measure: Number; unit: Percentage of subjects
Arm/Group | GSK257049 [5-17M] Group | GSK257049 [6-12W] Group | VeroRab Comparator [5-17M] Group | Menjugate Comparator [6-12W] Group
Number analyzed (Participants) | 4557 | 3996 | 2328 | 2007
Percentage of subjects
  ISA CD1 | 0.01 | 0.01 | 0.01 | 0.01
  MH CD1 | 0.05 | 0.04 | 0.09 | 0.05
  MH CD2 | 0.06 | 0.05 | 0.1 | 0.06

18. Secondary Outcome: Percentage of Subjects With Incident Severe Anaemia (ISA), Malaria Hospitalization (MH) and Fatal Malaria (FM) for Case Definitions (CD) Considered
Description: ISA CD considered were CD1, CD2 and CD3 (definitions mentioned in the previous outcome measure). MH CD considered were CD1 and CD2 (definitions mentioned in the previous outcome measure).FM CD considered were primary CD (PCD) and sedondary CDs 1 and 4 (SCD1 and SCD4). FM of PCD was defined as a case of severe malaria meeting the primary case definition of severe malaria disease with a fatal outcome. FM of SCD1 was defined as a case of severe malaria meeting the secondary case definition 1 severe malaria disease with a fatal outcome. FM of SCD4 was defined as a fatal case associated with International Classification Disease (ICD10) codes B50, B53 and/or B54. Code B50 corresponds to P. falciparum malaria including mixed infections of P. falciparum with any other Plasmodium species; Code B53 corresponds to other parasitologically confirmed malaria; Code B54 corresponds to unspecified malaria including clinically diagnosed malaria without parasitological confirmation.
Time Frame: From Month 2.5 to up to study end (with a median follow-up time post-Dose 1 of 48 months for 5-17M groups and 38 months for 6-12W groups)
Population: as for outcome 3
Measure: Number; unit: Percentage of subjects
Arm/Group | GSK257049 - GSK257049 [5-17M] Group | GSK257049 - Menjugate [5-17M] Group | VeroRab Comparator [5-17M] Group | GSK257049 -GSK257049 [6-12W] Group | GSK257049 - Menjugate [6-12W] Group | Menjugate Comparator [6-12W] Group
Number analyzed (Participants) | 2276 | 2306 | 2336 | 1985 | 2005 | 2007
Percentage of subjects
  ISA CD1 | 0.01 | 0.01 | 0.02 | 0.01 | 0.01 | 0.02
  ISA CD2 | 0.01 | 0.02 | 0.02 | 0.01 | 0.02 | 0.02
  ISA CD3 | 0.02 | 0.02 | 0.02 | 0.02 | 0.03 | 0.03
  MH CD1 | 0.07 | 0.1 | 0.12 | 0.06 | 0.07 | 0.08
  MH CD2 | 0.09 | 0.11 | 0.13 | 0.08 | 0.09 | 0.1
  FM PCD | 0 | 0 | 0 | 0 | 0 | 0
  FM SCD1 | 0 | 0 | 0 | 0 | 0 | 0
  FM SCD4 | 0 | 0 | 0 | 0 | 0.01 | 0

19. Secondary Outcome: Percentage of Subjects With Incident Severe Anaemia (ISA), Malaria Hospitalization (MH) and Fatal Malaria (FM) for Case Definitions (CD) Considered
Description: as for outcome 18
Time Frame: From Month 2.5 to Month 32
Population: as for outcome 3
Measure: Number; unit: Percentage of subjects
Arm/Group | GSK257049 - GSK257049 [5-17M] Group | GSK257049 - Menjugate [5-17M] Group | VeroRab Comparator [5-17M] Group | GSK257049 -GSK257049 [6-12W] Group | GSK257049 - Menjugate [6-12W] Group | Menjugate Comparator [6-12W] Group
Number analyzed (Participants) | 2276 | 2306 | 2336 | 1985 | 2005 | 2007
Percentage of subjects
  ISA CD1 | 0.01 | 0.01 | 0.01 | 0.1 | 0.01 | 0.01
  ISA CD2 | 0.01 | 0.01 | 0.02 | 0.01 | 0.01 | 0.01
  ISA CD3 | 0.01 | 0.02 | 0.02 | 0.02 | 0.02 | 0.02
  MH CD1 | 0.06 | 0.09 | 0.11 | 0.05 | 0.06 | 0.07
  MH CD2 | 0.08 | 0.1 | 0.12 | 0.07 | 0.08 | 0.09
  FM PCD | 0 | 0 | 0 | 0 | 0 | 0
  FM SCD1 | 0 | 0 | 0 | 0 | 0 | 0
  FM SCD4 | 0 | 0 | 0 | 0 | 0 | 0

20. Secondary Outcome: Percentage of Subjects With Prevalent Parasitemia, Prevalent Gametocytemia and Prevalent Severe and Moderate Anemia
Description: Prevalent parasitemia (PP) was defined as a documented P. falciparum asexual parasite density > 0 identified at timing of assessment. Prevalent gametocytemia (PG) was defined as a documented P. falciparum gametocyte density > 0 identified at a cross sectional survey. Prevalent severe anemia (PSA) was defined as a documented hemoglobin < 5.0 g/dL identified at timing of assessment. Prevalent moderate anemia (PMA) was defined as a documented hemoglobin < 8.0 g/dL identified at at timing of assessment. Results presented are uncorrected for the double enrollment of one subject receiving RTS,S/AS01.
Time Frame: At Month 20 (Booster)
Population: The analysis was performed on the ATP population for efficacy, which included all children who received all vaccinations according to protocol procedures and contributed to the time at risk in the follow-up period starting 14 days post Dose 3. Data was not collected for the participants in the 6-12W groups for the PG category.
Measure: Number; unit: Percentage of subjects
Arm/Group | GSK257049 [5-17M] Group | GSK257049 [6-12W] Group | VeroRab Comparator [5-17M] Group | Menjugate Comparator [6-12W] Group
Number analyzed (Participants) | 4140 | 3571 | 2100 | 1766
Percentage of subjects
  PP | 0.07 | 0.07 | 0.11 | 0.08
  PSA: number analyzed (Participants) | 4139 | 3571 | 2097 | 1765
  PSA | 0 | 0 | 0 | 0
  PMA: number analyzed (Participants) | 4139 | 3571 | 2097 | 1765
  PMA | 0.03 | 0.04 | 0.03 | 0.04
  PG: number analyzed (Participants) | 4021 | 0 | 2025 | 0
  PG | 0.03 |  | 0.04 |

21. Secondary Outcome: Percentage of Subjects With Prevalent Parasitemia and Prevalent Severe and Moderate Anemia
Description: Prevalent parasitemia (PP) was defined as a documented P. falciparum asexual parasite density > 0 identified at timing of assessment. Prevalent severe anemia (PSA) was defined as a documented hemoglobin < 5.0 g/dL identified at timing of assessment. Prevalent moderate anemia (PMA) was defined as a documented hemoglobin < 8.0 g/dL identified at timing of assessment. Analysis was performed on subjects aged 5-17 months at enrollment. Study End (Early) corresponds to children whose Month 32 visit took place after 30 June 2012 and who had one cross-sectional visit at study end. These children's last study visit was relatively earlier, with a median follow-up time of 14 months post Month 32. Study End (Late) corresponds to children whose Month 32 visit took place before (and including) 30 June 2012, and who had 2 cross-sectional visits after Month 32. These children's last study visit was relatively later, with a median follow-up time of 17 months post Month 32).
Time Frame: At Months 32, 44, at study end (median follow-up time of 48 months post-Dose 1 for 5-17 months age category and of 38 months post-Dose 1 for 6-12 weeks age category) (early and late)
Population: The analysis was performed on the ATP population for efficacy, which included all children who received all vaccinations according to protocol procedures and contributed to the time at risk in the follow-up period 14 days post Dose 3. Data was not collected for the participants in the 6-12W groups for the PP, PSA, PMA categories at M44, SE (Late).
Measure: Number; unit: Percentage of subjects
Arm/Group | GSK257049 - GSK257049 [5-17M] Group | GSK257049 - Menjugate [5-17M] Group | VeroRab Comparator [5-17M] Group | GSK257049 -GSK257049 [6-12W] Group | GSK257049 - Menjugate [6-12W] Group | Menjugate Comparator [6-12W] Group
Number analyzed (Participants) | 1935 | 1967 | 1979 | 1637 | 1656 | 1648
Percentage of subjects
  PP, Month 32: number analyzed (Participants) | 1935 | 1963 | 1976 | 1635 | 1656 | 1647
  PP, Month 32 | 0.09 | 0.1 | 0.14 | 0.09 | 0.11 | 0.1
  PSA, Month 32: number analyzed (Participants) | 1934 | 1967 | 1979 | 1637 | 1655 | 1648
  PSA, Month 32 | 0 | 0 | 0 | 0 | 0 | 0
  PMA, Month 32: number analyzed (Participants) | 1934 | 1967 | 1979 | 1637 | 1655 | 1648
  PMA, Month 32 | 0.02 | 0.02 | 0.02 | 0.02 | 0.04 | 0.03
  PP, Month 44: number analyzed (Participants) | 1039 | 1072 | 1093 | 0 | 0 | 0
  PP, Month 44 | 0.16 | 0.17 | 0.2 |  |  |
  PSA, Month 44: number analyzed (Participants) | 1041 | 1072 | 1094 | 0 | 0 | 0
  PSA, Month 44 | 0 | 0 | 0 |  |  |
  PMA, Month 44: number analyzed (Participants) | 1041 | 1072 | 1094 | 0 | 0 | 0
  PMA, Month 44 | 0.01 | 0.02 | 0.01 |  |  |
  PP, SE (Early): number analyzed (Participants) | 681 | 661 | 672 | 1481 | 1472 | 1487
  PP, SE (Early) | 0.09 | 0.1 | 0.14 | 0.11 | 0.14 | 0.13
  PSA, SE (Early): number analyzed (Participants) | 681 | 661 | 672 | 1481 | 1472 | 1486
  PSA, SE (Early) | 0 | 0 | 0 | 0 | 0 | 0
  PMA, SE (Early): number analyzed (Participants) | 681 | 661 | 672 | 1481 | 1472 | 1486
  PMA, SE (Early) | 0.01 | 0.02 | 0.03 | 0.03 | 0.03 | 0.03
  PP, SE (Late): number analyzed (Participants) | 1054 | 1059 | 1104 | 0 | 0 | 0
  PP, SE (Late) | 0.18 | 0.18 | 0.21 |  |  |
  PSA, SE (Late): number analyzed (Participants) | 1053 | 1057 | 1104 | 0 | 0 | 0
  PSA, SE (Late) | 0 | 0 | 0 |  |  |
  PMA, SE (Late): number analyzed (Participants) | 1053 | 1057 | 1104 | 0 | 0 | 0
  PMA, SE (Late) | 0.03 | 0.03 | 0.02 |  |  |

22. Secondary Outcome: Percentage of Subjects With Pneumonia, All-cause Hospitalization and Sepsis, as Per Case Definitions Assessed
Description: Pneumonia case definitions assessed are PCD and SCD 1, 2 and 3. Pneumonia of PCD was defined as cough or difficulty breathing AND tachypnea (≥ 50 breaths per minute < 1 year, ≥ 40 breaths per minute ≥ 1year) AND lower chest wall indrawing. Pneumonia of SCD1 was defined as pneumonia of PCD accompanied by chest X-ray (CXR) consolidation or pleural effusion on x-ray taken within 72 h of admission. Pneumonia of SCD2 was defined as pneumonia of PCD accompanied by consolidation or pleural effusion or other infiltrates on a chest x-ray taken within 72 h of admission. Pneumonia of SCD3 was defined as pneumonia of PCD accompanied by an oxygen saturation < 90%. All-cause hospitalization of PCD was defined as a medical hospitalization of any cause (excludes planned admissions for medical investigation/care or elective surgery and trauma). Sepsis cases were defined as a child with positive blood culture (CD1) or salmonella blood culture (CD2).
Time Frame: From Month 2.5 to Month 20
Population: as for outcome 3
Measure: Number; unit: Percentage of subjects
Arm/Group | GSK257049 [5-17M] Group | GSK257049 [6-12W] Group | VeroRab Comparator [5-17M] Group | Menjugate Comparator [6-12W] Group
Number analyzed (Participants) | 4557 | 3996 | 2328 | 2007
Percentage of subjects
  Pneumonia PCD | 0.03 | 0.04 | 0.03 | 0.04
  Pneumonia SCD1 | 0.01 | 0.01 | 0 | 0.01
  Pneumonia SCD2 | 0.02 | 0.03 | 0.02 | 0.03
  Pneumonia SCD3 | 0 | 0.01 | 0.01 | 0.01
  All-Cause Hospitalization PCD | 0.15 | 0.18 | 0.19 | 0.19
  Sepsis CD1 | 0.02 | 0.02 | 0.02 | 0.01
  Sepsis CD2 | 0.01 | 0.01 | 0.01 | 0.01

23. Secondary Outcome: Percentage of Subjects With Fatal Malaria (FM) and All-cause Mortality (ACM) as Per Case Definitions Assessed
Description: Fatal malaria case definitions assessed were PCD and SCD1. Fatal malaria of PCD was defined as a case of severe malaria meeting the primary case definition of severe malaria disease (defined in a previous outcome measure) with a fatal outcome. Fatal malaria of SCD1 was defined as a case of severe malaria meeting the secondary case definition 1 severe malaria disease (defined previously) with a fatal outcome. All-cause mortality case definitions assessed were the case definitions (CD) 1 and 2. All-cause mortality of CD1 was defined as a fatality (of any cause) (including mortality in the community and in hospital). All-cause mortality of CD2 was defined as a fatality (medical cause) (including mortality in the community and in hospital), at the exclusion of trauma which may be diagnosed by verbal autopsy. Results presented are uncorrected for double enrollment of one subject in 5-17 months age category receiving GSK257049 vaccine.
Time Frame: From Month 2.5 to Month 20
Population: as for outcome 3
Measure: Number; unit: Percentage of subjects
Arm/Group | GSK257049 [5-17M] Group | GSK257049 [6-12W] Group | VeroRab Comparator [5-17M] Group | Menjugate Comparator [6-12W] Group
Number analyzed (Participants) | 4557 | 3996 | 2328 | 2007
Percentage of subjects
  Fatal Malaria PCD | 0 | 0 | 0 | 0
  Fatal Malaria SCD1 | 0 | 0 | 0 | 0
  All-cause mortality CD1 | 0.01 | 0.01 | 0.01 | 0.01
  All-cause mortality CD2 | 0.01 | 0.01 | 0.01 | 0.01

24. Secondary Outcome: Percentage of Subjects With Pneumonia, All-cause Hospitalization/Mortality and Sepsis, as Per Case Definitions Assessed
Description: Pneumonia of PCD was defined as cough or difficulty breathing (on history) AND tachypnea (>= 50 breaths per minute < 1 year, >= 40 breaths per minute >= 1year) AND lower chest wall indrawing,SCD1 was defined as pneumonia of PCD accompanied by chest X-ray (CXR) consolidation or pleural effusion on x-ray taken within 72 h of admission,SCD2 was defined as pneumonia of PCD accompanied by consolidation or pleural effusion or other infiltrates on a chest x-ray taken within 72 h of admission,SCD3 was defined as pneumonia of PCD accompanied by an oxygen saturation less than 90%.All-cause hospitalization of PCD was defined as a medical hospitalization of any cause (excluding planned admissions for medical investigation/care or elective surgery and trauma).All-cause mortality of CD1 was defined as a fatality (of any cause),of CD2 defined as a fatality (medical cause).Sepsis of CD1 was defined as a child with positive blood culture;CD2 defined as a child with positive salmonella blood culture.
Time Frame: as for outcome 6
Population: as for outcome 3
Measure: Number; unit: Percentage of subjects
Arm/Group | GSK257049 - GSK257049 [5-17M] Group | GSK257049 - Menjugate [5-17M] Group | VeroRab Comparator [5-17M] Group | GSK257049 -GSK257049 [6-12W] Group | GSK257049 - Menjugate [6-12W] Group | Menjugate Comparator [6-12W] Group
Number analyzed (Participants) | 2276 | 2306 | 2336 | 1985 | 2005 | 2007
Percentage of subjects
  All-Cause Hospitalization PCD | 0.21 | 0.22 | 0.24 | 0.23 | 0.23 | 0.24
  Sepsis CD1 | 0.02 | 0.02 | 0.03 | 0.02 | 0.02 | 0.02
  Sepsis CD2 | 0.01 | 0.01 | 0.02 | 0.01 | 0.02 | 0.01
  Pneumonia PCD | 0.04 | 0.03 | 0.03 | 0.05 | 0.05 | 0.05
  Pneumonia SCD1 | 0.01 | 0.01 | 0.01 | 0.01 | 0.01 | 0.01
  Pneumonia SCD2 | 0.03 | 0.02 | 0.02 | 0.03 | 0.03 | 0.03
  Pneumonia SCD3 | 0 | 0 | 0.01 | 0.01 | 0.01 | 0.01
  All-Cause Mortality CD1 | 0.01 | 0.01 | 0.01 | 0.02 | 0.02 | 0.01
  All-Cause Mortality CD2 | 0.01 | 0.01 | 0.01 | 0.02 | 0.02 | 0.01

25. Secondary Outcome: Percentage of Subjects With Blood Transfusion, as Per Case Definition Assessed
Description: Blood transfusion case definition assessed was the case definition 1 (CD1). Blood transfusion of CD1 was defined as a child with inpatient admission with documented blood transfusion.
Time Frame: From Month 2.5 up to study end (median follow-up time of 48 months post-Dose 1 for 5-17 months age category and of 38 months post-Dose 1 for 6-12 weeks age category)
Population: as for outcome 3
Measure: Number; unit: Percentage of subjects
Arm/Group | GSK257049 - GSK257049 [5-17M] Group | GSK257049 - Menjugate [5-17M] Group | VeroRab Comparator [5-17M] Group | GSK257049 -GSK257049 [6-12W] Group | GSK257049 - Menjugate [6-12W] Group | Menjugate Comparator [6-12W] Group
Number analyzed (Participants) | 2276 | 2306 | 2336 | 1985 | 2005 | 2007
Percentage of subjects | 0.03 | 0.03 | 0.04 | 0.03 | 0.03 | 0.04

26. Secondary Outcome: Rate of All Episodes of Clinical P. Falciparum Malaria Infection (CPFMI) of Primary Case Definition (PCD), by Gender and Overall
Description: CPFMI of PCD = episode of malaria for which PFAP > 5000 parasites/µL accompanied by the presence of fever (axillary temperature ≥ 37.5°C at time of presentation) AND occurring in a child unwell brought for treatment to a healthcare facility OR a case of malaria meeting the PCD of severe malaria disease. Time to all episodes of CPFMI is expressed as a rate of all CPFMI (RaCPFMI), that is, person-year rate in each group (n/T). Analysis was performed on subjects aged 5-17 months and 6-12 weeks at enrollment. Results were presented by gender and overall.
Time Frame: From Month 2.5 to Month 32
Population: as for outcome 3
Measure: Number; unit: events per person-year
Arm/Group | GSK257049 - GSK257049 [5-17M] Group | GSK257049 - Menjugate [5-17M] Group | VeroRab Comparator [5-17M] Group | GSK257049 -GSK257049 [6-12W] Group | GSK257049 - Menjugate [6-12W] Group | Menjugate Comparator [6-12W] Group
Number analyzed (Participants) | 2276 | 2306 | 2336 | 1985 | 2005 | 2007
events per person-year
  PCD Females: number analyzed (Participants) | 1123 | 1137 | 1167 | 967 | 976 | 1014
  PCD Females | 0.72 | 0.8 | 1.11 | 0.76 | 0.79 | 1.06
  PCD Males: number analyzed (Participants) | 1153 | 1169 | 1169 | 1018 | 1029 | 993
  PCD Males | 0.65 | 0.81 | 1.19 | 0.83 | 0.96 | 1.01
  PCD Overall | 0.68 | 0.81 | 1.15 | 0.8 | 0.88 | 1.03

27. Secondary Outcome: Height, Weight and Mid Upper Arm Circumference for Age Z-score (HAZ, WAZ and MUACZ)
Description: Anthropometry consisted of length/height for age z-score [HAZ] (children < 2 years length measure and children ≥ 2 years standing height measure), weight for age z-score [WAZ] and mid-upper arm circumference for age z-score [MUACZ] measurements, where a HAZ < -1,5 z-score, indicates growth deficit, while a HAZ between -1,0 and ± 1,0 z-score, indicates normal height. A WAZ ≤ -3 z-score indicates a very low weight for age, a WAZ > -3 and ≤ -2 z-score indicates a low weight for age, a WAZ > - 2 z-score indicates normal weight. A MUACZ < -2 z-score indicates children that are wasted, a MUACZ < - 3 z-score indicates severely wasted children.
Time Frame: At Month 20 (Booster)
Population: The analysis was performed on the Intent-to-Treat (ITT) population, which included all children who received at least one dose of study vaccine.
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | GSK257049 [5-17M] Group | GSK257049 [6-12W] Group | VeroRab Comparator [5-17M] Group | Menjugate Comparator [6-12W] Group
Number analyzed (Participants) | 5948 | 4358 | 2974 | 2179
z-score
  HAZ: number analyzed (Participants) | 5048 | 4358 | 2974 | 2179
  HAZ | -1.6 (1) | -1.7 (1.1) | -1.6 (1) | -1.7 (1.2)
  WAZ | -1 (1) | -0.9 (1) | -1 (1) | -0.9 (1)
  MUACZ | -0.3 (0.9) | -0.1 (1) | -0.3 (0.9) | -0.1 (1)

28. Secondary Outcome: Height, Weight and Mid Upper Arm Circumference for Age Z-score (HAZ, WAZ and MUACZ)
Description: Anthropometry consisted of length/height for age z-score [HAZ] (children < 2 years length measure and children ≥ 2 years standing height measure), weight for age z-score [WAZ] and mid-upper arm circumference for age z-score [MUACZ] measurements, where a HAZ < -1,5 z-score, indicates growth deficit, while a HAZ between -1,0 and ± 1,0 z-score, indicates normal height. A WAZ ≤ -3 z-score indicates a very low weight for age, a WAZ > -3 and ≤ -2 z-score indicates a low weight for age, a WAZ > - 2 z-score indicates normal weight. A MUACZ < -2 z-score indicates children that are wasted, a MUACZ < - 3 z-score indicates severely wasted children. Note: The early study end refers to children whose last visit in the primary study phase (Month 32) was after 30 June 2012 and who by protocol had one cross-sectional study end and to late study end refers to children whose last visit in the primary study phase (Month 32) was after 30 June 2012 and who by protocol had one cross-sectional study end.
Time Frame: At Months 32, 44, at study end (early and late) (median follow-up time of 48 months post-Dose 1 for 5-17 months age category and of 38 months post-Dose 1 for 6-12 weeks age category)
Population: The analysis was performed on the ITT population, which included all children who received at least one dose of study vaccine. Data was not collected for the participants in the 6-12W groups for the HAZ, WAZ, MUACZ categories at Month 44 and at Study end Late time frames.
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | GSK257049 - GSK257049 [5-17M] Group | GSK257049 - Menjugate [5-17M] Group | VeroRab Comparator [5-17M] Group | GSK257049 -GSK257049 [6-12W] Group | GSK257049 - Menjugate [6-12W] Group | Menjugate Comparator [6-12W] Group
Number analyzed (Participants) | 2363 | 2382 | 2392 | 1726 | 1731 | 1725
z-score
  HAZ, Month 32 | -1.3 (1.0) | -1.4 (1.0) | -1.4 (1.0) | -1.5 (1.1) | -1.4 (1.1) | -1.5 (1.1)
  WAZ, Month 32 | -0.9 (0.9) | -1.0 (0.9) | -1.0 (0.9) | -0.9 (1.0) | -0.9 (1.0) | -0.9 (1.0)
  MUACZ, Month 32 | -0.4 (0.9) | -0.4 (0.9) | -0.4 (0.8) | -0.4 (0.9) | -0.3 (1.0) | -0.4 (1.0)
  HAZ, Month 44: number analyzed (Participants) | 1275 | 1289 | 1307 | 0 | 0 | 0
  HAZ, Month 44 | -1.1 (1.0) | -1.2 (0.9) | -1.2 (1.0) |  |  |
  WAZ, Month 44: number analyzed (Participants) | 1275 | 1289 | 1307 | 0 | 0 | 0
  WAZ, Month 44 | -0.9 (0.9) | -1.0 (0.9) | -0.9 (0.8) |  |  |
  MUACZ, Month 44: number analyzed (Participants) | 1275 | 1289 | 1307 | 0 | 0 | 0
  MUACZ, Month 44 | -0.7 (0.8) | -0.7 (0.9) | -0.6 (0.8) |  |  |
  HAZ, Study end Early: number analyzed (Participants) | 774 | 755 | 768 | 1555 | 1533 | 1549
  HAZ, Study end Early | -1.3 (1.0) | -1.3 (1.0) | -1.3 (1.0) | -1.4 (1.0) | -1.4 (1.0) | -1.4 (1.0)
  WAZ, Study end Early: number analyzed (Participants) | 774 | 755 | 768 | 1555 | 1533 | 1549
  WAZ, Study end Early | -1.0 (0.8) | -1.0 (0.8) | -1.0 (0.8) | -0.9 (0.9) | -0.9 (0.9) | -0.9 (0.9)
  MUACZ, Study end Early: number analyzed (Participants) | 774 | 755 | 768 | 1555 | 1533 | 1549
  MUACZ, Study end Early | -0.8 (0.9) | -0.8 (0.9) | -0.8 (0.8) | -0.5 (0.9) | -0.4 (0.9) | -0.5 (0.9)
  HAZ, Study end Late: number analyzed (Participants) | 1290 | 1283 | 1317 | 0 | 0 | 0
  HAZ, Study end Late | -1.0 (0.9) | -1.1 (0.9) | -1.1 (1.0) |  |  |
  WAZ, Study end Late: number analyzed (Participants) | 1290 | 1283 | 1317 | 0 | 0 | 0
  WAZ, Study end Late | -0.9 (0.9) | -1.0 (0.9) | -1.0 (0.8) |  |  |
  MUACZ, Study end Late: number analyzed (Participants) | 1290 | 1283 | 1317 | 0 | 0 | 0
  MUACZ, Study end Late | -0.7 (0.8) | -0.8 (0.9) | -0.7 (0.8) |  |  |

29. Secondary Outcome: Antibody Concentrations Against Plasmodium Falciparum Circumsporozoite (Anti-CS)
Description: Anti-CS antibody concentrations were determined by enzyme-linked immunosorbent assay (ELISA) and presented as geometric mean concentrations (GMCs), expressed in ELISA units per milliliter (EL.U/mL). The seropositivity cut-off for the endpoint was a GMC value ≥ 0.5 EL.U/mL. Results were assessed for the first 200 subjects enrolled in each study center.
Time Frame: At Day 0 and at Month 3
Population: The analysis was performed on the ATP population for immunogenicity, which included all first 200 children enrolled in each study center in each age category who received all vaccinations according to the protocol procedures.
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | GSK257049 [5-17M] Group | GSK257049 [6-12W] Group | VeroRab Comparator [5-17M] Group | Menjugate Comparator [6-12W] Group
Number analyzed (Participants) | 1036 | 1234 | 529 | 627
EL.U/mL
  Anti-CS, Day 0: number analyzed (Participants) | 1036 | 1234 | 526 | 627
  Anti-CS, Day 0 | 0.3 [0.3 to 0.3] | 0.4 [0.4 to 0.4] | 0.3 [0.3 to 0.3] | 0.4 [0.4 to 0.5]
  Anti-CS, Month 3: number analyzed (Participants) | 1034 | 1221 | 529 | 627
  Anti-CS, Month 3 | 621 [591.5 to 651.9] | 210.5 [198.2 to 223.6] | 0.3 [0.3 to 0.3] | 0.3 [0.3 to 0.3]

30. Secondary Outcome: Antibody Concentrations Against P. Falciparum Circumsporozoite (Anti-CS)
Description: Anti-CS antibody concentrations were determined by ELISA and presented as geometric mean concentrations (GMCs), expressed in EL.U/mL. The seropositivity cut-off for the endpoint was a GMC value ≥ 0.5 EL.U/mL. Results were assessed for the first 200 HIV-infected subjects enrolled in each study center. HIV infection was confirmed if present at screening or identified by morbidity surveillance, not infection confirmed by antibody testing after 18 months of age or by PCR, by the time of the analysis of results up to the Month 14 time point for the respective 5-17 months and 6-12 weeks age categories.
Time Frame: At Day 0 and at Month 3
Population: The analysis was performed on the HIV-ATP population for immunogenicity, which included all children included in the HIV-ITT population who received all vaccinations according to the protocol procedures.
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | GSK257049 [5-17M] Group | GSK257049 [6-12W] Group | VeroRab Comparator [5-17M] Group | Menjugate Comparator [6-12W] Group
Number analyzed (Participants) | 29 | 25 | 17 | 5
EL.U/mL
  Anti-CS, Day 0: number analyzed (Participants) | 28 | 25 | 16 | 5
  Anti-CS, Day 0 | 0.3 [0.2 to 0.5] | 0.3 [0.2 to 0.4] | 0.4 [0.3 to 0.5] | 0.3 [0.3 to 0.3]
  Anti-CS, Month 3: number analyzed (Participants) | 29 | 24 | 17 | 5
  Anti-CS, Month 3 | 264.7 [137.5 to 509.6] | 125.3 [58.1 to 270.3] | 0.5 [0.2 to 1.7] | 0.3 [0.3 to 0.3]

31. Secondary Outcome: Antibody Concentrations Against P. Falciparum Circumsporozoite (Anti-CS)
Description: Anti-CS antibody concentrations were determined by ELISA and presented as geometric mean concentrations (GMCs), expressed in EL.U/mL. The seropositivity cut-off for the endpoint was a GMC value ≥ 0.5 EL.U/mL.
Time Frame: At Months 20, 21 and 32
Population: The analysis was performed on the ATP population for immunogenicity, which included all first 200 children enrolled in each study center in each age category who received all vaccinations according to the protocol procedures. Data was not collected for the participants in the 5-17M groups for the Manhica site at any given time frame.
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | GSK257049 - GSK257049 [5-17M] Group | GSK257049 - Menjugate [5-17M] Group | VeroRab Comparator [5-17M] Group | GSK257049 -GSK257049 [6-12W] Group | GSK257049 - Menjugate [6-12W] Group | Menjugate Comparator [6-12W] Group
Number analyzed (Participants) | 442 | 438 | 426 | 530 | 569 | 554
EL.U/mL
  Anti-CS, Agogo - Month 20: number analyzed (Participants) | 55 | 57 | 54 | 55 | 55 | 66
  Anti-CS, Agogo - Month 20 | 34.1 [24.0 to 48.3] | 52.1 [41.3 to 65.7] | 0.3 [0.3 to 0.4] | 5.1 [3.4 to 7.6] | 5.6 [3.8 to 8.4] | 0.3 [0.2 to 0.3]
  Anti-CS, Agogo - Month 21: number analyzed (Participants) | 51 | 53 | 53 | 55 | 55 | 65
  Anti-CS, Agogo - Month 21 | 265.0 [220.9 to 317.9] | 48.3 [37.6 to 61.9] | 0.3 [0.2 to 0.3] | 137.6 [95.0 to 199.3] | 5.3 [3.5 to 8.0] | 0.3 [0.2 to 0.3]
  Anti-CS, Agogo - Month 32: number analyzed (Participants) | 53 | 54 | 54 | 52 | 53 | 64
  Anti-CS, Agogo - Month 32 | 46.3 [34.8 to 61.6] | 28.8 [21.8 to 37.9] | 0.3 [0.2 to 0.3] | 14.8 [9.5 to 23.1] | 2.9 [1.9 to 4.5] | 0.3 [0.3 to 0.4]
  Anti-CS, Bagamoyo - Month 20: number analyzed (Participants) | 16 | 18 | 25 | 47 | 54 | 42
  Anti-CS, Bagamoyo - Month 20 | 26.6 [14.2 to 49.9] | 23.1 [11.1 to 47.8] | 0.3 [0.3 to 0.3] | 6.9 [4.8 to 10.0] | 7.6 [5.1 to 11.4] | 0.3 [0.2 to 0.3]
  Anti-CS, Bagamoyo - Month 21: number analyzed (Participants) | 16 | 18 | 24 | 46 | 53 | 42
  Anti-CS, Bagamoyo - Month 21 | 306.6 [206.5 to 455.4] | 31.8 [19.4 to 52.2] | 0.6 [0.2 to 1.4] | 169.9 [129.8 to 222.5] | 7.2 [4.5 to 11.6] | 0.3 [0.2 to 0.4]
  Anti-CS, Bagamoyo - Month 32: number analyzed (Participants) | 16 | 17 | 24 | 43 | 49 | 40
  Anti-CS, Bagamoyo - Month 32 | 44.6 [27.2 to 73.3] | 16.9 [10.2 to 27.9] | 0.3 [0.3 to 0.3] | 14.4 [9.6 to 21.7] | 3.7 [2.4 to 5.7] | 0.3 [0.3 to 0.3]
  Anti-CS, Kilifi - Month 20: number analyzed (Participants) | 43 | 50 | 42 | 43 | 56 | 53
  Anti-CS, Kilifi - Month 20 | 34.3 [26.3 to 44.7] | 33.1 [26.3 to 41.6] | 0.3 [0.3 to 0.3] | 6.6 [4.6 to 9.6] | 6.1 [4.0 to 9.4] | 0.3 [0.2 to 0.3]
  Anti-CS, Kilifi - Month 21: number analyzed (Participants) | 40 | 49 | 41 | 41 | 54 | 51
  Anti-CS, Kilifi - Month 21 | 308.4 [251.8 to 377.7] | 24.3 [18.1 to 32.8] | 0.3 [0.3 to 0.3] | 229.3 [175.4 to 299.9] | 5.3 [3.4 to 8.2] | 0.3 [0.3 to 0.3]
  Anti-CS, Kilifi - Month 32: number analyzed (Participants) | 42 | 47 | 39 | 42 | 51 | 50
  Anti-CS, Kilifi - Month 32 | 59.4 [45.7 to 77.2] | 14.9 [11.0 to 20.2] | 0.3 [0.2 to 0.4] | 19.8 [14.1 to 27.8] | 2.8 [1.8 to 4.4] | 0.3 [0.3 to 0.3]
  Anti-CS, Kintampo - Month 20: number analyzed (Participants) | 57 | 51 | 52 | 52 | 55 | 46
  Anti-CS, Kintampo - Month 20 | 50.8 [37.2 to 69.5] | 36.6 [26.4 to 50.7] | 0.4 [0.3 to 0.5] | 3.8 [2.5 to 5.8] | 3.7 [2.5 to 5.6] | 0.3 [0.3 to 0.4]
  Anti-CS, Kintampo - Month 21: number analyzed (Participants) | 54 | 47 | 47 | 47 | 50 | 43
  Anti-CS, Kintampo - Month 21 | 266.8 [188.9 to 377.0] | 41.2 [31.2 to 54.6] | 0.3 [0.2 to 0.3] | 128.8 [95.7 to 173.4] | 3.2 [2.0 to 5.0] | 0.3 [0.3 to 0.4]
  Anti-CS, Kintampo - Month 32: number analyzed (Participants) | 50 | 46 | 49 | 47 | 47 | 42
  Anti-CS, Kintampo - Month 32 | 70.9 [55.2 to 90.9] | 20.2 [14.3 to 28.5] | 0.4 [0.3 to 0.5] | 13.3 [8.1 to 21.9] | 2.2 [1.4 to 3.4] | 0.3 [0.3 to 0.3]
  Anti-CS, Kombewa - Month 20: number analyzed (Participants) | 54 | 50 | 60 | 54 | 54 | 54
  Anti-CS, Kombewa - Month 20 | 39.8 [29.9 to 53.0] | 46.6 [33.2 to 65.3] | 0.3 [0.3 to 0.4] | 5.5 [3.6 to 8.4] | 8.7 [5.8 to 13.0] | 0.4 [0.3 to 0.5]
  Anti-CS, Kombewa - Month 21: number analyzed (Participants) | 52 | 50 | 59 | 50 | 51 | 52
  Anti-CS, Kombewa - Month 21 | 308.5 [252.4 to 377.0] | 37.1 [26.7 to 51.5] | 0.4 [0.3 to 0.4] | 146.3 [96.6 to 221.6] | 9.2 [6.0 to 14.2] | 0.4 [0.3 to 0.5]
  Anti-CS, Kombewa - Month 32: number analyzed (Participants) | 48 | 46 | 56 | 46 | 48 | 51
  Anti-CS, Kombewa - Month 32 | 53.8 [40.3 to 71.7] | 19.8 [14.1 to 27.7] | 0.3 [0.3 to 0.4] | 8.3 [4.8 to 14.3] | 4.3 [2.8 to 6.6] | 0.4 [0.3 to 0.4]
  Anti-CS, Korogwe - Month 20: number analyzed (Participants) | 55 | 61 | 52 | 52 | 48 | 57
  Anti-CS, Korogwe - Month 20 | 29.4 [21.4 to 40.4] | 28.2 [22.5 to 35.3] | 0.3 [0.3 to 0.3] | 7.9 [5.3 to 11.8] | 8.1 [5.2 to 12.7] | 0.3 [0.2 to 0.3]
  Anti-CS, Korogwe - Month 21: number analyzed (Participants) | 50 | 61 | 48 | 50 | 46 | 54
  Anti-CS, Korogwe - Month 21 | 305.6 [266.4 to 350.5] | 27.1 [20.7 to 35.5] | 0.3 [0.2 to 0.3] | 178.3 [141.2 to 225.1] | 7.6 [4.8 to 11.9] | 0.3 [0.2 to 0.4]
  Anti-CS, Korogwe - Month 32: number analyzed (Participants) | 52 | 56 | 44 | 49 | 42 | 48
  Anti-CS, Korogwe - Month 32 | 47.4 [37.5 to 59.9] | 16.8 [13.1 to 21.7] | 0.3 [0.2 to 0.3] | 19.6 [13.0 to 29.6] | 4.9 [3.0 to 7.9] | 0.3 [0.2 to 0.3]
  Anti-CS, Lambarene - Month 20: number analyzed (Participants) | 32 | 30 | 29 | 44 | 46 | 39
  Anti-CS, Lambarene - Month 20 | 8.2 [5.8 to 11.6] | 11.1 [7.0 to 17.6] | 0.3 [0.2 to 0.3] | 7.7 [5.1 to 11.6] | 8.3 [5.8 to 12.1] | 0.3 [0.3 to 0.3]
  Anti-CS, Lambarene - Month 21: number analyzed (Participants) | 32 | 30 | 29 | 43 | 45 | 35
  Anti-CS, Lambarene - Month 21 | 203.6 [155.1 to 267.3] | 10.6 [6.6 to 16.8] | 0.3 [0.2 to 0.3] | 251.3 [184.8 to 341.7] | 7.4 [5.0 to 10.8] | 0.3 [0.2 to 0.3]
  Anti-CS, Lambarene - Month 32: number analyzed (Participants) | 29 | 29 | 27 | 38 | 43 | 33
  Anti-CS, Lambarene - Month 32 | 23.0 [15.6 to 33.9] | 5.9 [3.6 to 9.9] | 0.3 [0.2 to 0.4] | 21.0 [13.9 to 31.7] | 4.1 [2.9 to 5.8] | 0.3 [0.2 to 0.3]
  Anti-CS, Lilongwe - Month 20: number analyzed (Participants) | 21 | 17 | 25 | 48 | 46 | 53
  Anti-CS, Lilongwe - Month 20 | 45.9 [28.6 to 73.8] | 22.2 [11.2 to 44.0] | 0.4 [0.2 to 0.7] | 5.1 [3.2 to 8.3] | 7.4 [4.7 to 11.5] | 0.3 [0.3 to 0.4]
  Anti-CS, Lilongwe - Month 21: number analyzed (Participants) | 23 | 15 | 24 | 44 | 45 | 51
  Anti-CS, Lilongwe - Month 21 | 285.0 [228.5 to 355.4] | 17.0 [8.1 to 35.7] | 0.3 [0.2 to 0.4] | 126.1 [92.7 to 171.5] | 8.0 [5.2 to 12.1] | 0.3 [0.2 to 0.4]
  Anti-CS, Lilongwe - Month 32: number analyzed (Participants) | 19 | 16 | 22 | 45 | 46 | 50
  Anti-CS, Lilongwe - Month 32 | 45.6 [28.8 to 72.3] | 12.7 [6.4 to 25.3] | 0.3 [0.2 to 0.4] | 15.4 [9.3 to 25.4] | 4.5 [3.1 to 6.6] | 0.3 [0.2 to 0.3]
  Anti-CS, Nanoro - Month 20: number analyzed (Participants) | 63 | 60 | 56 | 50 | 69 | 53
  Anti-CS, Nanoro - Month 20 | 57.2 [43.4 to 75.4] | 61.8 [46.3 to 82.4] | 0.3 [0.3 to 0.3] | 2.7 [1.7 to 4.4] | 3.2 [2.1 to 4.7] | 0.3 [0.3 to 0.4]
  Anti-CS, Nanoro - Month 21: number analyzed (Participants) | 63 | 60 | 56 | 50 | 68 | 53
  Anti-CS, Nanoro - Month 21 | 520.5 [443.4 to 611.1] | 71.1 [54.8 to 92.3] | 0.3 [0.2 to 0.3] | 163.2 [121.4 to 219.4] | 3.1 [2.0 to 4.6] | 0.3 [0.3 to 0.4]
  Anti-CS, Nanoro - Month 32: number analyzed (Participants) | 60 | 57 | 51 | 45 | 66 | 51
  Anti-CS, Nanoro - Month 32 | 69.2 [55.2 to 86.9] | 35.0 [25.7 to 47.9] | 0.3 [0.3 to 0.3] | 11.9 [7.4 to 19.2] | 2.8 [2.0 to 4.0] | 0.5 [0.4 to 0.6]
  Anti-CS, Siaya - Month 20: number analyzed (Participants) | 46 | 44 | 31 | 40 | 40 | 48
  Anti-CS, Siaya - Month 20 | 28.4 [18.4 to 44.0] | 32.8 [21.6 to 50.1] | 0.3 [0.3 to 0.4] | 7.0 [4.2 to 11.5] | 8.9 [5.5 to 14.2] | 0.4 [0.3 to 0.5]
  Anti-CS, Siaya - Month 21: number analyzed (Participants) | 45 | 42 | 28 | 41 | 39 | 45
  Anti-CS, Siaya - Month 21 | 398.1 [324.6 to 488.2] | 36.4 [22.6 to 58.6] | 0.3 [0.2 to 0.4] | 171.5 [109.8 to 267.9] | 8.4 [5.2 to 13.6] | 0.4 [0.3 to 0.5]
  Anti-CS, Siaya - Month 32: number analyzed (Participants) | 45 | 40 | 27 | 36 | 36 | 42
  Anti-CS, Siaya - Month 32 | 55.8 [41.4 to 75.3] | 21.7 [13.4 to 35.1] | 0.4 [0.3 to 0.5] | 23.6 [14.2 to 39.1] | 5.5 [3.3 to 9.2] | 0.5 [0.4 to 0.7]
  Anti-CS, Manhica - Month 20: number analyzed (Participants) | 0 | 0 | 0 | 45 | 46 | 43
  Anti-CS, Manhica - Month 20 |  |  |  | 12.3 [8.4 to 18.1] | 14.7 [10.0 to 21.5] | 0.3 [0.3 to 0.3]
  Anti-CS, Manhica - Month 21: number analyzed (Participants) | 0 | 0 | 0 | 36 | 38 | 28
  Anti-CS, Manhica - Month 21 |  |  |  | 260.2 [176.4 to 383.8] | 12.3 [7.7 to 19.5] | 0.3 [0.2 to 0.3]
  Anti-CS, Manhica - Month 32: number analyzed (Participants) | 0 | 0 | 0 | 35 | 34 | 30
  Anti-CS, Manhica - Month 32 |  |  |  | 25.4 [14.8 to 43.5] | 6.8 [4.0 to 11.5] | 0.3 [0.3 to 0.3]
  Anti-CS, Overall sites - Month 20 | 34.4 [30.7 to 38.6] | 35.4 [31.7 to 39.5] | 0.3 [0.3 to 0.3] | 5.9 [5.2 to 6.7] | 6.6 [5.8 to 7.5] | 0.3 [0.3 to 0.3]
  Anti-CS, Overall sites - Month 21: number analyzed (Participants) | 426 | 425 | 409 | 503 | 544 | 519
  Anti-CS, Overall sites - Month 21 | 318.2 [295.1 to 343.0] | 34.2 [30.5 to 38.3] | 0.3 [0.3 to 0.3] | 169.9 [153.8 to 187.7] | 6.2 [5.4 to 7.0] | 0.3 [0.3 to 0.3]
  Anti-CS, Overall sites - Month 32: number analyzed (Participants) | 414 | 408 | 393 | 478 | 515 | 501
  Anti-CS, Overall sites - Month 32 | 52.4 [47.8 to 57.6] | 19.3 [17.2 to 21.8] | 0.3 [0.3 to 0.3] | 15.9 [13.8 to 18.3] | 3.7 [3.3 to 4.2] | 0.3 [0.3 to 0.3]

32. Secondary Outcome: Antibody Concentrations Against P. Falciparum Circumsporozoite (Anti-CS)
Description: Anti-CS antibody concentrations were determined by ELISA and presented as geometric mean concentrations (GMCs), expressed in EL.U/mL. The seropositivity cut-off for the endpoint was a GMC value ≥ 0.5 EL.U/mL. Results for this endpoint were assessed for Agogo, Lilongwe and Siaya sites.
Time Frame: At Month 44 and at study end (median follow-up time of 48 months post-Dose 1 for 5-17 months age category and of 38 months post-Dose 1 for 6-12 weeks age category)
Population: The analysis was performed on the ATP population for immunogenicity, which included all first 200 children enrolled in each study center in each age category who received all vaccinations according to the protocol procedures. Data was not collected for the participants in the 6-12W groups at M44.
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | GSK257049 - GSK257049 [5-17M] Group | GSK257049 - Menjugate [5-17M] Group | VeroRab Comparator [5-17M] Group | GSK257049 -GSK257049 [6-12W] Group | GSK257049 - Menjugate [6-12W] Group | Menjugate Comparator [6-12W] Group
Number analyzed (Participants) | 104 | 101 | 98 | 101 | 103 | 131
EL.U/mL
  Anti-CS, Agogo - Month 44: number analyzed (Participants) | 47 | 50 | 45 | 0 | 0 | 0
  Anti-CS, Agogo - Month 44 | 27.7 [20.1 to 38.1] | 17.9 [13.5 to 23.6] | 0.3 [0.2 to 0.3] |  |  |
  Anti-CS, Agogo - Study end: number analyzed (Participants) | 47 | 48 | 49 | 32 | 35 | 51
  Anti-CS, Agogo - Study end | 23.2 [16.7 to 32.3] | 17.2 [12.7 to 23.3] | 0.3 [0.2 to 0.3] | 6.1 [3.2 to 11.4] | 2.1 [1.3 to 3.4] | 0.3 [0.2 to 0.4]
  Anti-CS, Lilongwe - Month 44: number analyzed (Participants) | 15 | 16 | 19 | 0 | 0 | 0
  Anti-CS, Lilongwe - Month 44 | 30.5 [21.4 to 43.5] | 8.5 [4.5 to 15.9] | 0.3 [0.2 to 0.3] |  |  |
  Anti-CS, Lilongwe - Study end: number analyzed (Participants) | 16 | 17 | 23 | 35 | 38 | 42
  Anti-CS, Lilongwe - Study end | 26.9 [18.3 to 39.5] | 7.2 [4.1 to 12.5] | 0.3 [0.3 to 0.3] | 10.9 [6.3 to 18.7] | 2.8 [1.8 to 4.2] | 0.3 [0.2 to 0.3]
  Anti-CS, Siaya - Month 44: number analyzed (Participants) | 41 | 35 | 22 | 0 | 0 | 0
  Anti-CS, Siaya - Month 44 | 41.4 [29.7 to 57.9] | 21.2 [14.0 to 32.0] | 0.5 [0.4 to 0.8] |  |  |
  Anti-CS, Siaya - Study end: number analyzed (Participants) | 41 | 34 | 26 | 34 | 30 | 38
  Anti-CS, Siaya - Study end | 27.4 [19.4 to 38.9] | 15.8 [10.2 to 24.4] | 0.4 [0.3 to 0.6] | 10.4 [6.1 to 17.7] | 3.3 [1.9 to 5.6] | 0.4 [0.3 to 0.6]
  Anti-CS, Overall - Month 44: number analyzed (Participants) | 103 | 101 | 86 | 0 | 0 | 0
  Anti-CS, Overall - Month 44 | 33.0 [26.9 to 40.3] | 16.8 [13.5 to 21.0] | 0.3 [0.3 to 0.4] |  |  |
  Anti-CS, Overall - Study end: number analyzed (Participants) | 104 | 99 | 98 | 101 | 103 | 131
  Anti-CS, Overall - Study end | 25.4 [20.6 to 31.2] | 14.4 [11.4 to 18.1] | 0.3 [0.3 to 0.4] | 8.9 [6.5 to 12.3] | 2.6 [2.0 to 3.4] | 0.3 [0.3 to 0.4]

33. Secondary Outcome: Antibody Concentrations Against P. Falciparum Circumsporozoite (Anti-CS), by Tertile
Description: Anti-CS antibody concentrations were determined by ELISA and presented as geometric mean concentrations (GMCs), expressed in EL.U/mL. The seropositivity cut-off for the endpoint was a GMC value ≥ 0.5 EL.U/mL. Results were presented by tertiles of anti-CS responses in the first 200 participants per site, based on subjects assessed for vaccine efficacy results.
Time Frame: At Month 3
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | GSK257049 - Menjugate [5-17M] Group | GSK257049 - Menjugate [6-12W] Group
Number analyzed (Participants) | 545 | 639
EL.U/mL
  Anti-CS, Tertile 1: number analyzed (Participants) | 181 | 212
  Anti-CS, Tertile 1 | 264.15 [238.2 to 292.9] | 78.45 [69.4 to 88.6]
  Anti-CS, Tertile 2: number analyzed (Participants) | 182 | 214
  Anti-CS, Tertile 2 | 613.79 [598.3 to 629.7] | 230.68 [224.7 to 236.8]
  Anti-CS, Tertile 3: number analyzed (Participants) | 182 | 213
  Anti-CS, Tertile 3 | 1351.41 [1276.3 to 1431] | 592.65 [557.8 to 629.6]
  Anti-CS, Across Tertiles | 603.77 [563.6 to 646.8] | 220.9 [204.1 to 239]

34. Secondary Outcome: Rate of All Episodes of Clinical P. Falciparum Malaria Infection (CPFMI) of Primary Case Definition (PCD), by Tertile
Description: CPFMI of PCD = episode of malaria for which PFAP > 5000 parasites/µL accompanied by presence of fever (axillary temperature ≥ 37.5°C at time of presentation) AND occurring in a child unwell brought for treatment to a healthcare facility OR a case of malaria meeting the PCD of severe malaria disease. Time to all episodes of CPFMI is expressed as a rate of all CPFMI (RaCPFMI), that is, person-year rate in each group (n/T). RaCPFMI was calculated by tertile of anti-CS response post primary vaccination pooled across sites, on subjects in GSK257049-Menjugate Groups (5-17M; 6-12W) and Comparator Groups (5-17M; 6-12W), taking into account the first 200 participants per site.
Time Frame: From Month 2.5 to Month 32
Population: as for outcome 3
Measure: Number; unit: events per person-year
Arm/Group | GSK257049 - Menjugate [5-17M] Group | VeroRab Comparator [5-17M] Group | GSK257049 - Menjugate [6-12W] Group | Menjugate Comparator [6-12W] Group
Number analyzed (Participants) | 182 | 565 | 214 | 677
events per person-year
  Tertile 1: number analyzed (Participants) | 181 | 565 | 212 | 677
  Tertile 1 | 0.68 | 1.21 | 1.29 | 0.93
  Tertile 2 | 0.78 | 1.21 | 0.7 | 0.93
  Tertile 3: number analyzed (Participants) | 182 | 565 | 213 | 677
  Tertile 3 | 1.03 | 1.21 | 0.58 | 0.93

35. Secondary Outcome: Antibody Concentrations Against P. Falciparum Circumsporozoite (Anti-CS), by Tertile
Description: as for outcome 33
Time Frame: At Month 21
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | GSK257049 - GSK257049 [5-17M] Group | GSK257049 -GSK257049 [6-12W] Group
Number analyzed (Participants) | 465 | 546
EL.U/mL
  Anti-CS, Tertile 1: number analyzed (Participants) | 154 | 181
  Anti-CS, Tertile 1 | 138.15 [123.5 to 154.5] | 47.99 [41.2 to 55.9]
  Anti-CS, Tertile 2: number analyzed (Participants) | 156 | 183
  Anti-CS, Tertile 2 | 311.35 [303.4 to 319.6] | 194.85 [189.9 to 200]
  Anti-CS, Tertile 3: number analyzed (Participants) | 155 | 182
  Anti-CS, Tertile 3 | 675.24 [632.8 to 720.5] | 479.44 [446.8 to 514.5]
  Anti-CS, Across Tertiles | 307.93 [286.2 to 331.3] | 165.31 [150 to 182.2]

36. Secondary Outcome: Rate of All Episodes of Clinical P. Falciparum Malaria Infection (CPFMI) of Primary Case Definition (PCD), by Tertile
Description: CPFMI of PCD = episode of malaria for which PFAP > 5000 parasites/µL accompanied by presence of fever (axillary temperature ≥ 37.5°C at time of presentation) AND occurring in a child unwell brought for treatment to a healthcare facility OR a case of malaria meeting the PCD of severe malaria disease. Time to all episodes of CPFMI is expressed as a rate of all CPFMI (RaCPFMI), that is, person-year rate in each group (n/T). RaCPFMI was calculated by tertile of anti-CS response post booster vaccination pooled across sites, on subjects in R3R (5-17M; 6-12W) (or R3R below) and C3C (5-17M; 6-12W) (or C3C below) groups taking into account the first 200 participants per site.
Time Frame: From Booster at Month 20 to Month 32
Population: as for outcome 3
Measure: Number; unit: events per person-year
Arm/Group | GSK257049 - GSK257049 [5-17M] Group | VeroRab Comparator [5-17M] Group | GSK257049 -GSK257049 [6-12W] Group | Menjugate Comparator [6-12W] Group
Number analyzed (Participants) | 156 | 479 | 420 | 594
events per person-year
  Tertile 1: number analyzed (Participants) | 154 | 479 | 420 | 594
  Tertile 1 | 0.68 | 1.21 | 0.99 | 0.94
  Tertile 2: number analyzed (Participants) | 156 | 479 | 362 | 594
  Tertile 2 | 0.68 | 1.21 | 0.84 | 0.94
  Tertile 3: number analyzed (Participants) | 155 | 479 | 276 | 594
  Tertile 3 | 0.77 | 1.21 | 0.64 | 0.94

37. Secondary Outcome: Antibody Concentrations Against Hepatitis B Surface Antigen (Anti-HBs)
Description: Antibody concentrations assessed by ELISA, were presented as geometric mean concentrations (GMCs), and expressed in milli-international units per milliliter (mIU/mL). The seropositivity and seroprotection cut-offs were ≥ 10 and 100 mIU/mL, respectively. Results were assessed for the first 200 subjects in each center.
Time Frame: At Day 0 and at Month 3
Population: The analysis was performed on the ATP population for immunogenicity, which included all first 200 children enrolled in each study center, for each age category who received all vaccinations according to the protocol procedures.
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | GSK257049 [5-17M] Group | GSK257049 [6-12W] Group | VeroRab Comparator [5-17M] Group | Menjugate Comparator [6-12W] Group
Number analyzed (Participants) | 1029 | 1213 | 526 | 627
mIU/mL
  Anti-HBs, Day 0: number analyzed (Participants) | 1017 | 1120 | 515 | 561
  Anti-HBs, Day 0 | 166.3 [148 to 186.8] | 8.6 [8 to 9.3] | 168.6 [142.8 to 199.2] | 8.5 [7.7 to 9.4]
  Anti-HBs, Month 3 | 81567.7 [75442.7 to 88189.9] | 13674.3 [12811.5 to 14595.3] | 127.5 [108.8 to 149.4] | 728.8 [643.6 to 825.2]

38. Secondary Outcome: Antibody Concentrations Against Hepatitis B Surface Antigen
Description: Antibody concentrations as assessed by ELISA, were presented as geometric mean concentrations (GMCs), and expressed in mIU/mL. The seropositivity and seroprotection cut-offs were ≥ 10 and 100 mIU/mL, respectively. Results were assessed for the first 200 HIV-infected subjects enrolled in each study center. HIV infection was confirmed if present at screening or identified by morbidity surveillance, not infection confirmed by antibody testing after 18 months of age or by PCR, by the time of the analysis of results up to the Month 14 time point for the respective 5-17 months and 6-12 weeks age categories.
Time Frame: At Day 0 and at Month 3
Population: as for outcome 30
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | GSK257049 [5-17M] Group | GSK257049 [6-12W] Group | VeroRab Comparator [5-17M] Group | Menjugate Comparator [6-12W] Group
Number analyzed (Participants) | 29 | 25 | 17 | 5
mIU/mL
  Anti-HBs, Day 0: number analyzed (Participants) | 28 | 25 | 15 | 5
  Anti-HBs, Day 0 | 98.6 [43.8 to 222] | 7.5 [4.8 to 11.6] | 63.6 [19.4 to 208.4] | 5 [5 to 5]
  Anti-HBs, Month 3: number analyzed (Participants) | 29 | 24 | 17 | 5
  Anti-HBs, Month 3 | 37476.5 [17766 to 79054.9] | 1996.2 [561.6 to 7095.8] | 37.1 [9.1 to 151.9] | 197.2 [7.7 to 5081.7]

39. Secondary Outcome: Antibody Concentrations Against Hepatitis B Surface Antigen (Anti-HBs)
Description: Antibody concentrations as assessed by ELISA, were presented as geometric mean concentrations (GMCs), and expressed in mIU/mL. The seropositivity and seroprotection cut-offs were ≥ 6.2 and 100 mIU/mL, respectively. Results were assessed for the first 200 subjects in each center.
Time Frame: At Months 20 and 21
Population: The analysis was performed on the ATP population for HBs immunogenicity post booster, which included the first 200 children enrolled in Korogwe, Lamberene and Lilongwe study centers in each age category who received the booster dose of GSK257049 vaccine and all vaccinations according to the protocol procedures.
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | GSK257049 - GSK257049 [5-17M] Group | GSK257049 -GSK257049 [6-12W] Group
Number analyzed (Participants) | 95 | 134
mIU/mL
  Anti-HBs, Month 20 | 5068.5 [3711.3 to 6922] | 1532.5 [1240.6 to 1893.2]
  Anti-HBs, Month 21: number analyzed (Participants) | 94 | 48
  Anti-HBs, Month 21 | 95206.4 [72395.4 to 125204.9] | 116458.1 [86865.7 to 156131.6]

40. Secondary Outcome: Antibody Titers Against Poliomyelitis (Anti-polio) Type 1, 2 and 3
Description: Anti-Polio 1, 2 and 3 antibody titers were presented as geometric mean titers (GMTs). The seroprotection cut-off for the assay was an antibody titer ≥ 1:8.
Time Frame: At Day 0 and at Month 3
Population: The ATP population for Polio Sabin™ immunogenicity included all subjects from the ATP population for immunogenicity (minus those who received ≥ 2 doses of Polio Sabin™ vaccine prior to Dose 1 of study vaccine, or who received at least one dose of a polio vaccine in co-administration with the study vaccine before one month post Dose 3 blood sample.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | GSK257049 [6-12W] Group | Menjugate Comparator [6-12W] Group
Number analyzed (Participants) | 931 | 474
Titer
  Anti-Polio 1, Day 0: number analyzed (Participants) | 928 | 469
  Anti-Polio 1, Day 0 | 47.4 [41.7 to 53.8] | 43.3 [36.2 to 51.9]
  Anti-Polio 1, Month 3: number analyzed (Participants) | 913 | 464
  Anti-Polio 1, Month 3 | 334.9 [295.2 to 379.8] | 417.6 [351.4 to 496.2]
  Anti-Polio 2, Day 0: number analyzed (Participants) | 928 | 468
  Anti-Polio 2, Day 0 | 38.6 [34.6 to 43.2] | 40.3 [34.2 to 47.5]
  Anti-Polio 2, Month 3: number analyzed (Participants) | 913 | 466
  Anti-Polio 2, Month 3 | 372.1 [334.5 to 414.0] | 450.8 [393.9 to 516.0]
  Anti-Polio 3, Day 0 | 9.4 [8.6 to 10.3] | 9.1 [8.0 to 10.3]
  Anti-Polio 3, Month 3: number analyzed (Participants) | 913 | 466
  Anti-Polio 3, Month 3 | 80.0 [71.0 to 90.1] | 95.9 [82.0 to 112.2]

41. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms
Description: Assessed solicited local symptoms included pain, redness and swelling. Any = the incidence of a particular symptom, regardless of intensity grade. Grade 3 pain = cried when limb was moved, spontaneously painful. Grade 3 redness/swelling = redness/swelling spreading beyond 20 millimeters (mm) of injection site.
Time Frame: During the 7-day (Days 0-6) post-primary vaccination period following each dose and across doses
Population: The analysis was performed on the ITT population, which included all children who received at least one dose of study vaccine and had their symptom sheets filled in.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK257049 [5-17M] Group | VeroRab Comparator [5-17M] Group | GSK257049 [6-12W] Group | Menjugate Comparator [6-12W] Group
Number analyzed (Participants) | 1479 | 721 | 1462 | 738
Participants
  Any Pain, Dose 1 | 247 | 61 | 435 | 215
  Grade 3 Pain, Dose 1 | 0 | 0 | 10 | 7
  Any Redness, Dose 1 | 66 | 26 | 176 | 89
  Grade 3 Redness, Dose 1 | 2 | 0 | 3 | 3
  Any Swelling, Dose 1 | 140 | 77 | 227 | 125
  Grade 3 Swelling, Dose 1 | 6 | 0 | 27 | 29
  Any Pain, Dose 2: number analyzed (Participants) | 1435 | 708 | 1412 | 721
  Any Pain, Dose 2 | 179 | 41 | 383 | 178
  Grade 3 Pain, Dose 2: number analyzed (Participants) | 1435 | 708 | 1412 | 721
  Grade 3 Pain, Dose 2 | 3 | 0 | 5 | 3
  Any Redness, Dose 2: number analyzed (Participants) | 1435 | 708 | 1412 | 721
  Any Redness, Dose 2 | 26 | 18 | 124 | 90
  Grade 3 Redness, Dose 2: number analyzed (Participants) | 1435 | 708 | 1412 | 721
  Grade 3 Redness, Dose 2 | 3 | 0 | 3 | 1
  Any Swelling, Dose 2: number analyzed (Participants) | 1435 | 708 | 1412 | 721
  Any Swelling, Dose 2 | 140 | 50 | 228 | 128
  Grade 3 Swelling, Dose 2: number analyzed (Participants) | 1435 | 708 | 1412 | 721
  Grade 3 Swelling, Dose 2 | 15 | 0 | 29 | 17
  Any Pain, Dose 3: number analyzed (Participants) | 1407 | 699 | 1378 | 710
  Any Pain, Dose 3 | 108 | 22 | 345 | 153
  Grade 3 Pain, Dose 3: number analyzed (Participants) | 1407 | 699 | 1378 | 710
  Grade 3 Pain, Dose 3 | 0 | 0 | 8 | 2
  Any Redness, Dose 3: number analyzed (Participants) | 1407 | 699 | 1378 | 710
  Any Redness, Dose 3 | 42 | 13 | 113 | 63
  Grade 3 Redness, Dose 3: number analyzed (Participants) | 1407 | 699 | 1378 | 710
  Grade 3 Redness, Dose 3 | 2 | 0 | 1 | 1
  Any Swelling, Dose 3: number analyzed (Participants) | 1407 | 699 | 1378 | 710
  Any Swelling, Dose 3 | 134 | 35 | 185 | 111
  Grade 3 Swelling, Dose 3: number analyzed (Participants) | 1407 | 699 | 1378 | 710
  Grade 3 Swelling, Dose 3 | 9 | 0 | 9 | 12
  Any Pain, Across doses | 401 | 105 | 705 | 342
  Grade 3 Pain, Across doses | 3 | 0 | 23 | 12
  Any Redness, Across doses | 122 | 49 | 292 | 163
  Grade 3 Redness, Across doses | 6 | 0 | 7 | 5
  Any Swelling, Across doses | 303 | 119 | 427 | 248
  Grade 3 Swelling, Across doses | 25 | 0 | 59 | 53

42. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms
Description: Assessed solicited general symptoms were drowsiness, irritability, loss of appetite, fever [defined as axillary temperature equal to or above (≥) 37.5 degrees Celsius (°C)]. Any = occurrence of the symptom regardless of intensity grade or relationship to vaccination. Grade 3 symptom = symptom that prevented normal activity. Grade 3 fever = fever > 39.0 °C. Related = symptom assessed by the investigator as related to the vaccination.
Time Frame: During the 7-day (Days 0-6) post-primary vaccination period following each dose and across doses
Population: as for outcome 41
Measure: Count of Participants; unit: Participants
Arm/Group | GSK257049 [5-17M] Group | GSK257049 [6-12W] Group | VeroRab Comparator [5-17M] Group | Menjugate Comparator [6-12W] Group
Number analyzed (Participants) | 1479 | 1462 | 721 | 738
Participants
  Any Drowsiness, Dose 1 | 91 | 164 | 27 | 65
  Grade 3 Drowsiness, Dose 1 | 3 | 1 | 0 | 1
  Related Drowsiness, Dose 1 | 33 | 88 | 8 | 26
  Any Irritability, Dose 1 | 165 | 370 | 41 | 157
  Grade 3 Irritability, Dose 1 | 0 | 10 | 0 | 3
  Related Irritability, Dose 1 | 64 | 226 | 16 | 84
  Any Loss of appetite, Dose 1 | 202 | 124 | 71 | 52
  Grade 3 Loss of appetite, Dose 1 | 3 | 2 | 0 | 0
  Related Loss of appetite, Dose 1 | 71 | 67 | 24 | 24
  Any Fever, Dose 1 | 385 | 459 | 108 | 192
  Grade 3 Fever, Dose 1 | 29 | 5 | 7 | 2
  Related Fever, Dose 1 | 200 | 326 | 52 | 127
  Any Drowsiness, Dose 2: number analyzed (Participants) | 1435 | 1412 | 708 | 721
  Any Drowsiness, Dose 2 | 99 | 135 | 37 | 55
  Grade 3 Drowsiness, Dose 2: number analyzed (Participants) | 1435 | 1412 | 708 | 721
  Grade 3 Drowsiness, Dose 2 | 1 | 0 | 0 | 0
  Related Drowsiness, Dose 2: number analyzed (Participants) | 1435 | 1412 | 708 | 721
  Related Drowsiness, Dose 2 | 61 | 74 | 26 | 15
  Any Irritability, Dose 2: number analyzed (Participants) | 1435 | 1412 | 708 | 721
  Any Irritability, Dose 2 | 192 | 289 | 45 | 123
  Grade 3 Irritability, Dose 2: number analyzed (Participants) | 1435 | 1412 | 708 | 721
  Grade 3 Irritability, Dose 2 | 2 | 7 | 0 | 0
  Related Irritability, Dose 2: number analyzed (Participants) | 1435 | 1412 | 708 | 721
  Related Irritability, Dose 2 | 114 | 175 | 28 | 57
  Any Loss of appetite, Dose 2: number analyzed (Participants) | 1435 | 1412 | 708 | 721
  Any Loss of appetite, Dose 2 | 151 | 105 | 47 | 43
  Grade 3 Loss of appetite, Dose 2: number analyzed (Participants) | 1435 | 1412 | 708 | 721
  Grade 3 Loss of appetite, Dose 2 | 0 | 0 | 0 | 0
  Related Loss of appetite, Dose 2: number analyzed (Participants) | 1435 | 1412 | 708 | 721
  Related Loss of appetite, Dose 2 | 89 | 60 | 24 | 8
  Any Fever, Dose 2: number analyzed (Participants) | 1435 | 1412 | 708 | 721
  Any Fever, Dose 2 | 503 | 411 | 100 | 154
  Grade 3 Fever, Dose 2: number analyzed (Participants) | 1435 | 1412 | 708 | 721
  Grade 3 Fever, Dose 2 | 42 | 9 | 10 | 6
  Related Fever, Dose 2: number analyzed (Participants) | 1435 | 1412 | 708 | 721
  Related Fever, Dose 2 | 267 | 278 | 42 | 89
  Any Drowsiness, Dose 3: number analyzed (Participants) | 1407 | 1378 | 699 | 710
  Any Drowsiness, Dose 3 | 97 | 124 | 29 | 44
  Grade 3 Drowsiness, Dose 3: number analyzed (Participants) | 1407 | 1378 | 699 | 710
  Grade 3 Drowsiness, Dose 3 | 1 | 1 | 0 | 1
  Related Drowsiness, Dose 3: number analyzed (Participants) | 1407 | 1378 | 699 | 710
  Related Drowsiness, Dose 3 | 52 | 49 | 16 | 19
  Any Irritability, Dose 3: number analyzed (Participants) | 1407 | 1378 | 699 | 710
  Any Irritability, Dose 3 | 138 | 287 | 27 | 104
  Grade 3 Irritability, Dose 3: number analyzed (Participants) | 1407 | 1378 | 699 | 710
  Grade 3 Irritability, Dose 3 | 1 | 3 | 0 | 2
  Related Irritability, Dose 3: number analyzed (Participants) | 1407 | 1378 | 699 | 710
  Related Irritability, Dose 3 | 76 | 144 | 15 | 54
  Any Loss of appetite, Dose 3: number analyzed (Participants) | 1407 | 1378 | 699 | 710
  Any Loss of appetite, Dose 3 | 138 | 106 | 40 | 45
  Grade 3 Loss of appetite, Dose 3: number analyzed (Participants) | 1407 | 1378 | 699 | 710
  Grade 3 Loss of appetite, Dose 3 | 2 | 0 | 0 | 1
  Related Loss of appetite, Dose 3: number analyzed (Participants) | 1407 | 1378 | 699 | 710
  Related Loss of appetite, Dose 3 | 76 | 44 | 18 | 20
  Any Fever, Dose 3: number analyzed (Participants) | 1407 | 1378 | 699 | 710
  Any Fever, Dose 3 | 457 | 429 | 77 | 111
  Grade 3 Fever, Dose 3: number analyzed (Participants) | 1407 | 1378 | 699 | 710
  Grade 3 Fever, Dose 3 | 39 | 13 | 7 | 3
  Related Fever, Dose 3: number analyzed (Participants) | 1407 | 1378 | 699 | 710
  Related Fever, Dose 3 | 262 | 280 | 32 | 57
  Any Drowsiness, Across doses | 230 | 285 | 78 | 121
  Grade 3 Drowsiness, Across doses | 5 | 2 | 0 | 2
  Related Drowsiness, Across doses | 121 | 144 | 44 | 51
  Any Irritability, Across doses | 369 | 574 | 96 | 244
  Grade 3 Irritability, Across doses | 3 | 17 | 0 | 5
  Related Irritability, Across doses | 207 | 363 | 54 | 139
  Any Loss of appetite, Across doses | 398 | 243 | 132 | 104
  Grade 3 Loss of appetite, Across doses | 5 | 2 | 0 | 1
  Related Loss of appetite, Across doses | 206 | 128 | 61 | 41
  Any Fever, Across doses | 897 | 839 | 235 | 331
  Grade 3 Fever, Across doses | 105 | 26 | 24 | 11
  Related Fever, Across doses | 547 | 598 | 110 | 209

43. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms
Description: as for outcome 41
Time Frame: During the 7-day (Days 0-6) post-booster vaccination period
Population: The analysis was performed on the ITT population, which included all children who received at least one dose of study vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK257049 - GSK257049 [5-17M] Group | GSK257049 - Menjugate [5-17M] Group | VeroRab Comparator [5-17M] Group | GSK257049 -GSK257049 [6-12W] Group | GSK257049 - Menjugate [6-12W] Group | Menjugate Comparator [6-12W] Group
Number analyzed (Participants) | 641 | 639 | 633 | 608 | 625 | 621
Participants
  Any Pain | 109 | 45 | 41 | 59 | 29 | 25
  Grade 3 Pain | 0 | 0 | 0 | 0 | 0 | 0
  Any Redness | 15 | 13 | 8 | 9 | 12 | 9
  Grade 3 Redness | 3 | 0 | 0 | 1 | 0 | 0
  Any Swelling | 42 | 35 | 30 | 45 | 28 | 43
  Grade 3 Swelling | 9 | 1 | 0 | 5 | 0 | 2

44. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms
Description: as for outcome 42
Time Frame: During the 7-day (Days 0-6) post-booster vaccination period
Population: as for outcome 43
Measure: Count of Participants; unit: Participants
Arm/Group | GSK257049 - GSK257049 [5-17M] Group | GSK257049 - Menjugate [5-17M] Group | VeroRab Comparator [5-17M] Group | GSK257049 -GSK257049 [6-12W] Group | GSK257049 - Menjugate [6-12W] Group | Menjugate Comparator [6-12W] Group
Number analyzed (Participants) | 641 | 639 | 633 | 608 | 625 | 621
Participants
  Any Drowsiness | 55 | 22 | 21 | 33 | 19 | 15
  Grade 3 Drowsiness | 1 | 0 | 0 | 0 | 0 | 0
  Related Drowsiness | 34 | 10 | 13 | 19 | 6 | 5
  Any Irritability | 63 | 25 | 18 | 46 | 23 | 23
  Grade 3 Irritability | 1 | 0 | 0 | 0 | 0 | 0
  Related Irritability | 40 | 12 | 8 | 27 | 10 | 6
  Any Loss of appetite | 66 | 27 | 21 | 45 | 27 | 18
  Grade 3 Loss of appetite | 1 | 0 | 0 | 0 | 0 | 0
  Related Loss of appetite | 39 | 14 | 13 | 26 | 8 | 6
  Any Fever | 233 | 70 | 45 | 152 | 52 | 58
  Grade 3 Fever | 34 | 6 | 5 | 9 | 7 | 10
  Related Fever | 151 | 29 | 16 | 80 | 15 | 18

45. Secondary Outcome: Number of Doses With Seizures by Diagnostic Certainty Level
Description: Diagnostic certainty levels included: Level 1- Witnessed sudden loss of consciousness and generalized, tonic, clonic, tonic-clonic, or atonic motor manifestations; Level 2- History of unconsciousness and generalized, tonic, clonic, tonic-clonic, or atonic motor manifestations; Level 3- History of unconsciousness and other generalized motor manifestations; Level 4- Reported generalized convulsive seizure with insufficient evidence to meet the case definition; Level 5- Not a case of generalized convulsive seizure.
Time Frame: During the 7-day (Days 0-6) post-booster vaccination period, at Month 20 + 7 Day (Days 0-6)
Population: as for outcome 43
Measure: Number; unit: Doses
Arm/Group | GSK257049 - GSK257049 [5-17M] Group | GSK257049 - Menjugate [5-17M] Group | VeroRab Comparator [5-17M] Group | GSK257049 -GSK257049 [6-12W] Group | GSK257049 - Menjugate [6-12W] Group | Menjugate Comparator [6-12W] Group
Number analyzed (Participants) | 2447 | 2472 | 2473 | 1825 | 1837 | 1827
Doses
  Level 1 | 1 | 1 | 0 | 1 | 0 | 0
  Level 2 | 5 | 2 | 1 | 3 | 0 | 1
  Level 3 | 0 | 0 | 0 | 0 | 0 | 0
  Level 4 | 1 | 0 | 0 | 0 | 0 | 0
  Level 5 | 1 | 1 | 0 | 0 | 0 | 0

46. Secondary Outcome: Number of Subjects Reporting Mucocutaneous Changes (All Levels)
Description: Levels of mucocutaneous changes reported were: cutaneous and mucosal change; cutaneous only change; mucosal only change; cutaneous change focused on the nappy/diaper area. Mucocutaneous changes results calculated based on the first 200 subjects in the 6-12 weeks age category in each study center were enrolled, and with available data (i.e. who received a booster dose).
Time Frame: During the 30-day (Days 0-29) post-booster vaccination
Population: as for outcome 43
Measure: Count of Participants; unit: Participants
Arm/Group | GSK257049 -GSK257049 [6-12W] Group | GSK257049 - Menjugate [6-12W] Group | Menjugate Comparator [6-12W] Group
Number analyzed (Participants) | 605 | 617 | 614
Participants | 64 | 47 | 59

47. Secondary Outcome: Number of Subjects Reporting Any Meningitis and Encephalitis Serious Adverse Events (SAEs)
Description: Meningitis and encephalitis SAEs included: meningitis/encephalitis; meningitis/encephalitis viral; meningism; meningitis haemophilus; meningitis meningococcal; meningitis pneumococcal; meningitis tuberculous; encephalomyelitis.
Time Frame: At Month 0 until study end (median follow-up time of 48 months post-Dose 1 for 5-17 months age category and of 38 months post-Dose 1 for 6-12 weeks age category)
Population: as for outcome 43
Measure: Count of Participants; unit: Participants
Arm/Group | GSK257049 - GSK257049 [5-17M] Group | GSK257049 - Menjugate [5-17M] Group | VeroRab Comparator [5-17M] Group | GSK257049 -GSK257049 [6-12W] Group | GSK257049 - Menjugate [6-12W] Group | Menjugate Comparator [6-12W] Group
Number analyzed (Participants) | 2976 | 2972 | 2974 | 2180 | 2178 | 2179
Participants | 15 | 12 | 5 | 7 | 8 | 7

48. Secondary Outcome: Number of Subjects Reporting Any Meningitis and Encephalitis SAEs
Description: Meningitis and encephalitis SAEs included: meningitis/encephalitis; meningitis haemophilus; meningitis meningococcal; meningitis tuberculous; encephalomyelitis.
Time Frame: From Booster up to study end (median follow-up time of 48 months post-Dose 1 for 5-17 months age category and of 38 months post-Dose 1 for 6-12 weeks age category)
Population: as for outcome 43
Measure: Count of Participants; unit: Participants
Arm/Group | GSK257049 - GSK257049 [5-17M] Group | GSK257049 - Menjugate [5-17M] Group | VeroRab Comparator [5-17M] Group | GSK257049 -GSK257049 [6-12W] Group | GSK257049 - Menjugate [6-12W] Group | Menjugate Comparator [6-12W] Group
Number analyzed (Participants) | 2681 | 2719 | 2702 | 1966 | 1996 | 1976
Participants | 4 | 4 | 0 | 0 | 2 | 3

49. Secondary Outcome: Number of Subjects Reporting Any Potential Immune-mediated Disorders (pIMDs)
Description: Potential immune-mediated diseases (pIMDs) are a subset of AEs that include autoimmune diseases and other inflammatory and/or neurologic disorders of interest which may or may not have an autoimmune aetiology.
Time Frame: From Month 0 up to study end (median follow-up time of 48 months post-Dose 1 for 5-17 months age category and of 38 months post-Dose 1 for 6-12 weeks age category)
Population: as for outcome 43
Measure: Count of Participants; unit: Participants
Arm/Group | GSK257049 - GSK257049 [5-17M] Group | GSK257049 - Menjugate [5-17M] Group | VeroRab Comparator [5-17M] Group | GSK257049 -GSK257049 [6-12W] Group | GSK257049 - Menjugate [6-12W] Group | Menjugate Comparator [6-12W] Group
Number analyzed (Participants) | 2976 | 2972 | 2974 | 2180 | 2178 | 2179
Participants | 5 | 1 | 4 | 3 | 1 | 2

50. Secondary Outcome: Number of Subjects With Any Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination. Unsolicited AEs were calculated based on the first 200 subjects enrolled in each study center.
Time Frame: Within the 30-day (Days 0-29) post-primary vaccination period
Population: as for outcome 43
Measure: Count of Participants; unit: Participants
Arm/Group | GSK257049 [5-17M] Group | GSK257049 [6-12W] Group | VeroRab Comparator [5-17M] Group | Menjugate Comparator [6-12W] Group
Number analyzed (Participants) | 1479 | 1462 | 721 | 738
Participants | 1273 | 1161 | 626 | 600

51. Secondary Outcome: Number of Subjects With Unsolicited AEs Related to or Leading to Vaccination Withdrawal
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Related = AE assessed by the investigator as related to the vaccination. Unsolicited AEs were calculated based on the first 200 subjects enrolled in each study center.
Time Frame: Within the 30-day (Days 0-29) post-primary vaccination period
Population: as for outcome 43
Measure: Count of Participants; unit: Participants
Arm/Group | GSK257049 [5-17M] Group | GSK257049 [6-12W] Group | VeroRab Comparator [5-17M] Group | Menjugate Comparator [6-12W] Group
Number analyzed (Participants) | 3997 | 4358 | 2003 | 2179
Participants | 399 | 578 | 72 | 231

52. Secondary Outcome: Number of Subjects With Any Unsolicited AEs
Description: as for outcome 50
Time Frame: Within the 30-day (days 0-29) post-booster vaccination period
Population: as for outcome 43
Measure: Count of Participants; unit: Participants
Arm/Group | GSK257049 - GSK257049 [5-17M] Group | GSK257049 - Menjugate [5-17M] Group | VeroRab Comparator [5-17M] Group | GSK257049 -GSK257049 [6-12W] Group | GSK257049 - Menjugate [6-12W] Group | Menjugate Comparator [6-12W] Group
Number analyzed (Participants) | 641 | 639 | 633 | 608 | 625 | 621
Participants | 232 | 205 | 215 | 231 | 239 | 240

53. Secondary Outcome: Number of Subjects With Unsolicited AEs Related to or Leading to Vaccination Withdrawal
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Related = AE assessed by the investigator as related to the vaccination. Unsolicited AEs were calculated based on the subgroup of the first 200 subjects enrolled in each study center, who were reported with HIV infected status ((HIV status either as per general medical history taken at screening or as identified by morbidity surveillance).
Time Frame: Within the 30-day (Days 0-29) post-primary and post-booster vaccination period in HIV-infected children
Population: The analysis was performed on the HIV-ITT population, which included all children who received at least one dose of GSK257049 vaccine and were identified as HIV-infected, that is, confirmed to be HIV-infected via identification as positive for HIV by Polymerase Chain Reaction (PCR), or by antibody at 18 months or older.
Measure: Count of Participants; unit: Participants
Groups:
- GSK257049 Group: Pooled group between GSK257049 [5-17M] Group and GSK257049 [6-12W] Group.
- GSK257049 -GSK257049 Group: Pooled group between GSK257049 -GSK257049 [5-17M] Group and GSK257049 -GSK257049 [6-12W] Group.
- GSK257049 - Menjugate Group: Pooled group between GSK257049 - Menjugate [5-17M] Group and GSK257049 - Menjugate [6-12W] Group.
- Comparator Group: Pooled Group between VeroRab Comparator [5-17M] Group and Menjugate Comparator [6-12W] Group.
Arm/Group | GSK257049 Group | GSK257049 -GSK257049 Group | GSK257049 - Menjugate Group | Comparator Group
Number analyzed (Participants) | 84 | 33 | 35 | 41
Participants
  Any AE(s), post-primary vaccination: number analyzed (Participants) | 84 | 0 | 0 | 41
  Any AE(s), post-primary vaccination | 13 | 0 | 0 | 3
  Any AE(s), post-booster vaccination: number analyzed (Participants) | 0 | 33 | 35 | 28
  Any AE(s), post-booster vaccination | 0 | 2 | 0 | 0

54. Secondary Outcome: Number of Subjects With Unsolicited AEs Related to or Leading to Vaccination Withdrawal in the Low-weight (LW) and Very Low-weight (VLW) Category
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Related = AE assessed by the investigator as related to the vaccination. Unsolicited AEs were calculated based on the subgroup of the first 200 subjects enrolled in each study center, who were reported with HIV infected status ((HIV status either as per general medical history taken at screening or as identified by morbidity surveillance). Low-weight subjects were defined as subjects whose weight for age z-score (WAZ) was > -3 and ≤ -2. Very low-weight subjects were defined as subjects whose weight for age z-score (WAZ) was ≤ -3.
Time Frame: Within the 30-day (Days 0-29) post-primary vaccination period in HIV-infected children
Population: The analysis was performed on the HIV-ITT population, which included low-weight and very low-weight children who received at least one dose of GSK257049 vaccine and were identified as HIV-infected, that is, confirmed to be HIV-infected via identification as positive for HIV by Polymerase Chain Reaction (PCR), or by antibody at 18 months or older.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK257049 [5-17M] Group | GSK257049 [6-12W] Group | VeroRab Comparator [5-17M] Group | Menjugate Comparator [6-12W] Group
Number analyzed (Participants) | 695 | 221 | 364 | 126
Participants
  Any AE(s), in LW | 68 | 38 | 21 | 17
  Any AE(s), in VLW: number analyzed (Participants) | 207 | 147 | 97 | 67
  Any AE(s), in VLW | 27 | 24 | 6 | 10

55. Secondary Outcome: Number of Subjects With Unsolicited AEs Related to Vaccination in the Low-weight (LW) and Very Low-weight (VLW) Category
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Related = AE assessed by the investigator as related to the vaccination. Unsolicited AEs were calculated based on the subgroup of the first 200 subjects enrolled in each study center. Low-weight subjects were defined as subjects whose weight for age z-score (WAZ) was > -3 and ≤ -2. Very low-weight subjects were defined as subjects whose weight for age z-score (WAZ) was ≤ -3.
Time Frame: Within the 30-day (Days 0-29) post-booster vaccination period
Population: The analysis was performed on a subset of subjects from the ITT population, which included low-weight (LW) and very low-weight (VLW) children who received at least one dose of study vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK257049 - GSK257049 [5-17M] Group | GSK257049 - Menjugate [5-17M] Group | VeroRab Comparator [5-17M] Group | GSK257049 -GSK257049 [6-12W] Group | GSK257049 - Menjugate [6-12W] Group | Menjugate Comparator [6-12W] Group
Number analyzed (Participants) | 273 | 297 | 293 | 230 | 208 | 195
Participants
  Any AE(s) in LW | 4 | 1 | 0 | 2 | 0 | 0
  Any AE(s) in VLW: number analyzed (Participants) | 48 | 49 | 59 | 45 | 45 | 68
  Any AE(s) in VLW | 5 | 0 | 1 | 2 | 0 | 1

56. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: From Month 0 up to Month 14
Population: as for outcome 43
Measure: Count of Participants; unit: Participants
Arm/Group | GSK257049 [5-17M] Group | GSK257049 [6-12W] Group | VeroRab Comparator [5-17M] Group | Menjugate Comparator [6-12W] Group
Number analyzed (Participants) | 5948 | 4358 | 2974 | 2179
Participants | 1040 | 782 | 634 | 419

57. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: as for outcome 56
Time Frame: During the 30-day (Days 0-29) post-primary vaccination period
Population: as for outcome 43
Measure: Count of Participants; unit: Participants
Arm/Group | GSK257049 [5-17M] Group | GSK257049 [6-12W] Group | VeroRab Comparator [5-17M] Group | Menjugate Comparator [6-12W] Group
Number analyzed (Participants) | 5948 | 4358 | 2974 | 2179
Participants | 312 | 192 | 181 | 96

58. Secondary Outcome: Number of Subjects With Serious Adversee Events (SAEs)
Description: as for outcome 56
Time Frame: From Month 0 up to Month 20
Population: as for outcome 43
Measure: Count of Participants; unit: Participants
Arm/Group | GSK257049 [5-17M] Group | GSK257049 [6-12W] Group | VeroRab Comparator [5-17M] Group | Menjugate Comparator [6-12W] Group
Number analyzed (Participants) | 5948 | 4358 | 2974 | 2179
Participants | 1108 | 959 | 676 | 503

59. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: as for outcome 56
Time Frame: From Booster (at Month 20) up to study end (median follow-up time of 48 months post-Dose 1 for 5-17 months age category and of 38 months post-Dose 1 for 6-12 weeks age category)
Population: as for outcome 43
Measure: Count of Participants; unit: Participants
Arm/Group | GSK257049 - GSK257049 [5-17M] Group | GSK257049 - Menjugate [5-17M] Group | VeroRab Comparator [5-17M] Group | GSK257049 -GSK257049 [6-12W] Group | GSK257049 - Menjugate [6-12W] Group | Menjugate Comparator [6-12W] Group
Number analyzed (Participants) | 2681 | 2719 | 2702 | 1966 | 1996 | 1976
Participants | 276 | 316 | 287 | 180 | 193 | 201

60. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: as for outcome 56
Time Frame: as for outcome 49
Population: The analysis was performed, across age categories for which groups were pooled from the ITT population, which included all children who received at least one dose of study vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK257049 - GSK257049 [5-17M] Group | GSK257049 - Menjugate [5-17M] Group | VeroRab Comparator [5-17M] Group | GSK257049 -GSK257049 [6-12W] Group | GSK257049 - Menjugate [6-12W] Group | Menjugate Comparator [6-12W] Group
Number analyzed (Participants) | 2976 | 2972 | 2974 | 2180 | 2178 | 2179
Participants | 720 | 752 | 846 | 580 | 602 | 619

61. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: as for outcome 56
Time Frame: Within the 30-day (Days 0-29) post-booster vaccination period
Population: as for outcome 43
Measure: Count of Participants; unit: Participants
Arm/Group | GSK257049 - GSK257049 [5-17M] Group | GSK257049 - Menjugate [5-17M] Group | VeroRab Comparator [5-17M] Group | GSK257049 -GSK257049 [6-12W] Group | GSK257049 - Menjugate [6-12W] Group | Menjugate Comparator [6-12W] Group
Number analyzed (Participants) | 2447 | 2472 | 2473 | 1825 | 1837 | 1827
Participants | 34 | 22 | 27 | 19 | 19 | 20

62. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: as for outcome 56
Time Frame: From Month 0 up to Booster (Month 20), from Month 0 up to study end and from Month 20 up to study end
Population: The analysis was performed on a subset of subjects from the ITT population, which included all children who received at least one dose of study vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK257049 -GSK257049 Group | GSK257049 - Menjugate Group | Comparator Group
Number analyzed (Participants) | 51 | 54 | 48
Participants
  Any SAE(s), Month 0 - Month 20 | 43 | 39 | 36
  Any SAE(s), Month 0 - Study end | 47 | 46 | 42
  Any SAE(s), Month 20 - Study end: number analyzed (Participants) | 38 | 42 | 32
  Any SAE(s), Month 20 - Study end | 19 | 19 | 16

63. Secondary Outcome: Number of Low-weight (LW) Subjects With Serious Adverse Events (SAEs)
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity. Low-weight subjects were defined as subjects whose weight for age z-score (WAZ) was > -3 and ≤ -2.
Time Frame: From Month 0 up to Month 20
Population: The analysis was performed on the ITT population, which included low weight (LW) children who received at least one dose of study vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK257049 [5-17M] Group | GSK257049 [6-12W] Group | VeroRab Comparator [5-17M] Group | Menjugate Comparator [6-12W] Group
Number analyzed (Participants) | 695 | 221 | 364 | 126
Participants | 174 | 63 | 89 | 38

64. Secondary Outcome: Number of Low-weight (LW) Subjects With Serious Adverse Events (SAEs)
Description: as for outcome 63
Time Frame: From Booster (Month 20) up to study end (median follow-up time of 48 months post-Dose 1 for 5-17 months age category and of 38 months post-Dose 1 for 6-12 weeks age category)
Population: The analysis was performed on a subset of subjects from the ITT population, which included low weight (LW) children who received at least one dose of study vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK257049 - GSK257049 [5-17M] Group | GSK257049 - Menjugate [5-17M] Group | VeroRab Comparator [5-17M] Group | GSK257049 -GSK257049 [6-12W] Group | GSK257049 - Menjugate [6-12W] Group | Menjugate Comparator [6-12W] Group
Number analyzed (Participants) | 277 | 304 | 297 | 232 | 211 | 195
Participants | 32 | 40 | 38 | 34 | 21 | 24

65. Secondary Outcome: Number of Very Low-weight (VLW) Subjects With Serious Adverse Events (SAEs)
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity. Very low-weight subjects were defined as subjects whose weight for age z-score (WAZ) was ≤ -3.
Time Frame: From Month 0 up to Month 20
Population: The analysis was performed on a subset of subjects from the ITT population, which included very-low weight (VLW) children who received at least one dose of study vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK257049 [5-17M] Group | GSK257049 [6-12W] Group | VeroRab Comparator [5-17M] Group | Menjugate Comparator [6-12W] Group
Number analyzed (Participants) | 207 | 147 | 97 | 67
Participants | 55 | 48 | 28 | 17

66. Secondary Outcome: Number of Very Low-weight Subjects With Serious Adverse Events (SAEs)
Description: as for outcome 65
Time Frame: From Booster (Month 20) up to study end (median follow-up time of 48 months post-Dose 1 for 5-17 months age category and of 38 months post-Dose 1 for 6-12 weeks age category)]
Population: as for outcome 65
Measure: Count of Participants; unit: Participants
Arm/Group | GSK257049 - GSK257049 [5-17M] Group | GSK257049 - Menjugate [5-17M] Group | VeroRab Comparator [5-17M] Group | GSK257049 -GSK257049 [6-12W] Group | GSK257049 - Menjugate [6-12W] Group | Menjugate Comparator [6-12W] Group
Number analyzed (Participants) | 48 | 50 | 60 | 48 | 47 | 68
Participants | 5 | 8 | 11 | 6 | 9 | 15

67. Secondary Outcome: Number of Subjects With Fatal Outcomes, by Gender
Description: Mortality was presented as overall mortality (up to Month 20 and up to study end), mortality due to severe malaria as per secondary case definition(SCD), cerebral malaria as per secondary case definition (SCD), meningitis, fatal all-cause traumas and fatal malaria. SCD= Plasmodium falciparum malaria > 5000 parasites/mcL and 1 or more markers of severe malaria (prostration, respiratory distress, Blantyre score ≤ 2, seizures 2 or more, hypoglycemia < 2.2 mmol/L, acidosis BE ≤ -10.0 mmol/L,lactate ≥ 5.0 mmol/L, anemia < 5.0 g/dL.
Time Frame: From Month 0 up to study end (SE - median follow-up time of 48 months post-Dose 1 for 5-17 months age category and of 38 months post-Dose 1 for 6-12 weeks age category)
Population: as for outcome 43
Measure: Count of Participants; unit: Participants
Arm/Group | GSK257049 - GSK257049 [5-17M] Group | GSK257049 - Menjugate [5-17M] Group | VeroRab Comparator [5-17M] Group | GSK257049 -GSK257049 [6-12W] Group | GSK257049 - Menjugate [6-12W] Group | Menjugate Comparator [6-12W] Group
Number analyzed (Participants) | 1509 | 1500 | 1503 | 1116 | 1118 | 1100
Participants
  Overall Mortality (M0-M20), Females: number analyzed (Participants) | 1467 | 1500 | 1503 | 1064 | 1060 | 1100
  Overall Mortality (M0-M20), Females | 27 | 20 | 14 | 20 | 24 | 13
  Overall Mortality (M0-SE), Females: number analyzed (Participants) | 1467 | 1500 | 1503 | 1064 | 1060 | 1100
  Overall Mortality (M0-SE), Females | 35 | 32 | 17 | 27 | 29 | 16
  Overall Mortality (M0-M20), Males: number analyzed (Participants) | 1509 | 1472 | 1471 | 1116 | 1118 | 1079
  Overall Mortality (M0-M20), Males | 19 | 8 | 19 | 20 | 20 | 21
  Overall Mortality (M0-SE), Males: number analyzed (Participants) | 1509 | 1472 | 1471 | 1116 | 1118 | 1079
  Overall Mortality (M0-SE), Males | 26 | 19 | 29 | 24 | 26 | 26
  Severe Malaria SCD, All, Females: number analyzed (Participants) | 1467 | 1500 | 1503 | 1064 | 1060 | 1100
  Severe Malaria SCD, All, Females | 75 | 107 | 100 | 57 | 49 | 75
  Severe Malaria SCD, All, Males: number analyzed (Participants) | 1509 | 1472 | 1471 | 1116 | 1118 | 1079
  Severe Malaria SCD, All, Males | 87 | 115 | 134 | 78 | 80 | 79
  Severe Malaria SCD, Fatal, Females: number analyzed (Participants) | 1467 | 1500 | 1503 | 1064 | 1060 | 1100
  Severe Malaria SCD, Fatal, Females | 4 | 4 | 2 | 2 | 0 | 0
  Severe Malaria SCD, Fatal, Males: number analyzed (Participants) | 1509 | 1472 | 1471 | 1116 | 1118 | 1079
  Severe Malaria SCD, Fatal, Males | 3 | 4 | 2 | 2 | 2 | 2
  Cerebral Malaria SCD, All, Females: number analyzed (Participants) | 1467 | 1500 | 1503 | 1064 | 1060 | 1100
  Cerebral Malaria SCD, All, Females | 16 | 14 | 7 | 1 | 5 | 7
  Cerebral Malaria SCD, All, Males: number analyzed (Participants) | 1509 | 1472 | 1471 | 1116 | 1118 | 1079
  Cerebral Malaria SCD, All, Males | 10 | 14 | 9 | 9 | 7 | 3
  Cerebral Malaria SCD, Fatal, Females: number analyzed (Participants) | 1467 | 1500 | 1503 | 1064 | 1060 | 1100
  Cerebral Malaria SCD, Fatal, Females | 3 | 4 | 2 | 1 | 0 | 0
  Cerebral Malaria SCD, Fatal, Males: number analyzed (Participants) | 1509 | 1472 | 1471 | 1116 | 1118 | 1079
  Cerebral Malaria SCD, Fatal, Males | 2 | 1 | 0 | 1 | 1 | 0
  Meningitis, All, Females: number analyzed (Participants) | 1467 | 1500 | 1503 | 1064 | 1060 | 1100
  Meningitis, All, Females | 5 | 5 | 1 | 2 | 2 | 3
  Meningitis, All, Males: number analyzed (Participants) | 1509 | 1472 | 1471 | 1116 | 1118 | 1079
  Meningitis, All, Males | 6 | 5 | 2 | 3 | 5 | 3
  Meningitis, Fatal, Females: number analyzed (Participants) | 1467 | 1500 | 1503 | 1064 | 1060 | 1100
  Meningitis, Fatal, Females | 2 | 3 | 0 | 0 | 0 | 1
  Meningitis, Fatal, Males: number analyzed (Participants) | 1509 | 1472 | 1471 | 1116 | 1118 | 1079
  Meningitis, Fatal, Males | 2 | 0 | 1 | 1 | 1 | 2
  Fatal All-Cause Traumas, Females: number analyzed (Participants) | 1467 | 1500 | 1503 | 1064 | 1060 | 1100
  Fatal All-Cause Traumas, Females | 3 | 4 | 1 | 1 | 1 | 2
  Fatal All-Cause Traumas, Males: number analyzed (Participants) | 1509 | 1472 | 1471 | 1116 | 1118 | 1079
  Fatal All-Cause Traumas, Males | 4 | 1 | 3 | 1 | 2 | 0
  Fatal Malaria, Females: number analyzed (Participants) | 1467 | 1500 | 1503 | 1064 | 1060 | 1100
  Fatal Malaria, Females | 9 | 8 | 4 | 5 | 4 | 3
  Fatal Malaria, Males: number analyzed (Participants) | 1509 | 1472 | 1471 | 1116 | 1118 | 1079
  Fatal Malaria, Males | 4 | 9 | 8 | 3 | 8 | 3

ADVERSE EVENTS:
Time Frame: Solicited local and general symptoms: during the 7-day (Days 0-6) post-vaccination periods; Unsolicited AEs: during the 30-day (Days 0-29) post-vaccination periods; SAEs: from Day 0 up to study end (median follow-up of 48 months for 5-17M subjects and of 38 months for 6-12W subjects).
Arm/Group | GSK257049 [5-17M] Group | GSK257049 [6-12W] Group | VeroRab Comparator [5-17M] Group | Menjugate Comparator [6-12W] Group
All-Cause Mortality (participants affected / at risk) | 112/5948 | 46/4358 | 106/2974 | 42/2179
Serious Adverse Events (participants affected / at risk) | 1475/5948 | 1186/4358 | 848/2974 | 622/2179
Other Adverse Events (participants affected / at risk) | 1410/1479 | 1360/1462 | 664/721 | 691/738
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK257049 [5-17M] Group (N=5948) | GSK257049 [6-12W] Group (N=4358) | VeroRab Comparator [5-17M] Group (N=2974) | Menjugate Comparator [6-12W] Group (N=2179)
Anaemia (Blood and lymphatic system disorders) | 277 (329) | 198 (258) | 198 (246) | 116 (138)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemolysis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Hypochromic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intravascular haemolysis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Leukaemoid reaction (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymphadenitis (Blood and lymphatic system disorders) | 7 (7) | 1 (1) | 1 (1) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial septal defect (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebral palsy (Congenital, familial and genetic disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Choledochal cyst (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Congenital megacolon (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Cryptorchism (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fallot's tetralogy (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Glucose-6-phosphate dehydrogenase deficiency (Congenital, familial and genetic disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Hydrocele (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Phimosis (Congenital, familial and genetic disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Sickle cell anaemia (Congenital, familial and genetic disorders) | 5 (5) | 4 (4) | 1 (1) | 5 (5)
Sickle cell anaemia with crisis (Congenital, familial and genetic disorders) | 8 (15) | 5 (10) | 6 (8) | 5 (10)
Trisomy 21 (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urethral valves (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ventricular septal defect (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Deafness (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hearing impaired (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Periorbital oedema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aphthous stomatitis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Enteritis (Gastrointestinal disorders) | 28 (28) | 17 (17) | 15 (15) | 18 (18)
Food poisoning (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Gastritis (Gastrointestinal disorders) | 2 (2) | 3 (3) | 2 (2) | 4 (4)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal motility disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ileus paralytic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Inguinal hernia, obstructive (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 2 (3) | 0 (0) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intussusception (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rectal polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rectal prolapse (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Stress ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Umbilical hernia, obstructive (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Death (General disorders) | 4 (4) | 3 (3) | 0 (0) | 3 (3)
Drowning (General disorders) | 5 (5) | 1 (1) | 3 (3) | 1 (1)
Generalised oedema (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hernia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypothermia (General disorders) | 2 (2) | 2 (2) | 0 (0) | 1 (1)
Injection site reaction (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 28 (28) | 27 (27) | 16 (16) | 18 (18)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Hepatitis acute (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hepatitis toxic (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Allergy to arthropod sting (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Immune reconstitution inflammatory syndrome (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abscess (Infections and infestations) | 14 (14) | 12 (12) | 5 (5) | 5 (5)
Abscess jaw (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abscess limb (Infections and infestations) | 1 (1) | 1 (1) | 3 (3) | 1 (1)
Abscess neck (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acarodermatitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Aids dementia complex (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Amoebiasis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Arthritis bacterial (Infections and infestations) | 9 (9) | 6 (6) | 1 (1) | 1 (1)
Ascariasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atypical pneumonia (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Bacterial infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Bone tuberculosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Brain abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Breast abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchiolitis (Infections and infestations) | 38 (42) | 32 (33) | 18 (24) | 24 (26)
Bronchitis (Infections and infestations) | 28 (31) | 17 (18) | 21 (22) | 3 (3)
Bronchopneumonia (Infections and infestations) | 68 (76) | 54 (60) | 40 (42) | 34 (36)
Bullous impetigo (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Burkholderia cepacia complex sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Burn infection (Infections and infestations) | 3 (3) | 1 (1) | 0 (0) | 1 (1)
Candida infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 15 (15) | 10 (10) | 6 (6) | 6 (6)
Cellulitis of male external genital organ (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cellulitis orbital (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cellulitis pharyngeal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Central nervous system viral infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebral malaria (Infections and infestations) | 8 (8) | 2 (3) | 0 (0) | 2 (2)
Cholera (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 6 (6) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis bacterial (Infections and infestations) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Croup infectious (Infections and infestations) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Dermatitis infected (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Disseminated tuberculosis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dysentery (Infections and infestations) | 24 (24) | 10 (10) | 9 (9) | 7 (7)
Eczema infected (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Empyema (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Encephalitis (Infections and infestations) | 5 (5) | 1 (1) | 2 (2) | 1 (1)
Encephalitis viral (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Encephalomyelitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Enterococcal sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Erysipelas (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Escherichia sepsis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Escherichia urinary tract infection (Infections and infestations) | 1 (1) | 3 (3) | 2 (2) | 2 (2)
Exanthema subitum (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Febrile infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Furuncle (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 302 (335) | 333 (379) | 177 (192) | 171 (192)
Gastroenteritis escherichia coli (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis salmonella (Infections and infestations) | 5 (5) | 7 (7) | 0 (0) | 4 (4)
Gastroenteritis shigella (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal candidiasis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Giardiasis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Gingivitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Groin abscess (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Haemophilus sepsis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Helminthic infection (Infections and infestations) | 10 (12) | 3 (3) | 6 (6) | 1 (1)
Hepatitis a (Infections and infestations) | 4 (4) | 0 (0) | 1 (1) | 1 (1)
Hepatitis b (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatitis infectious (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hiv associated nephropathy (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hiv infection (Infections and infestations) | 41 (41) | 36 (36) | 18 (18) | 12 (12)
Hiv infection who clinical stage ii (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hiv infection who clinical stage iii (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hiv infection who clinical stage iv (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Impetigo (Infections and infestations) | 3 (3) | 4 (4) | 3 (3) | 1 (1)
Infected skin ulcer (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Klebsiella sepsis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Laryngitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Listeria sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Liver abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lobar pneumonia (Infections and infestations) | 11 (11) | 17 (18) | 7 (8) | 7 (8)
Lower respiratory tract infection (Infections and infestations) | 5 (5) | 4 (4) | 6 (6) | 2 (2)
Ludwig angina (Infections and infestations) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Lymph node abscess (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Lymph node tuberculosis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Lymphadenitis bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malaria (Infections and infestations) | 639 (850) | 392 (525) | 423 (533) | 236 (303)
Mastoiditis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Measles (Infections and infestations) | 9 (9) | 24 (24) | 5 (5) | 8 (8)
Meningitis (Infections and infestations) | 10 (10) | 5 (5) | 1 (1) | 3 (3)
Meningitis haemophilus (Infections and infestations) | 3 (3) | 1 (1) | 0 (0) | 1 (1)
Meningitis meningococcal (Infections and infestations) | 5 (5) | 0 (0) | 0 (0) | 1 (1)
Meningitis pneumococcal (Infections and infestations) | 1 (1) | 3 (3) | 0 (0) | 2 (2)
Meningitis salmonella (Infections and infestations) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Meningitis tuberculous (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Meningitis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Moraxella infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mumps (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mycobacterium ulcerans infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 10 (10) | 3 (3) | 4 (5) | 1 (1)
Oropharyngeal candidiasis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 5 (5) | 2 (2) | 3 (3) | 2 (2)
Otitis externa (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 29 (29) | 22 (22) | 22 (22) | 7 (7)
Otitis media acute (Infections and infestations) | 4 (4) | 3 (3) | 2 (2) | 1 (1)
Otitis media chronic (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Parotitis (Infections and infestations) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Perineal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Periorbital cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Peritonitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Plasmodium ovale infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumococcal bacteraemia (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pneumococcal sepsis (Infections and infestations) | 9 (9) | 9 (10) | 3 (3) | 3 (3)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 2 (2) | 5 (5) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 417 (532) | 424 (547) | 223 (287) | 202 (286)
Pneumonia pneumococcal (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pneumonia streptococcal (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pneumonia viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Postoperative wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pseudomonal sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 8 (9) | 12 (12) | 4 (4) | 2 (2)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyoderma (Infections and infestations) | 2 (2) | 0 (0) | 3 (3) | 0 (0)
Pyomyositis (Infections and infestations) | 2 (2) | 2 (2) | 3 (3) | 0 (0)
Rabies (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 4 (4) | 1 (1) | 2 (2) | 0 (0)
Rubella (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Salmonella bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Salmonella sepsis (Infections and infestations) | 70 (73) | 60 (63) | 42 (42) | 37 (40)
Salmonellosis (Infections and infestations) | 4 (4) | 0 (0) | 2 (2) | 0 (0)
Schistosomiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 60 (61) | 38 (38) | 43 (46) | 13 (15)
Septic shock (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Shigella infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin bacterial infection (Infections and infestations) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Skin infection (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 9 (10) | 10 (10) | 1 (1) | 2 (2)
Staphylococcal skin infection (Infections and infestations) | 3 (3) | 1 (1) | 2 (2) | 1 (1)
Streptococcal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Streptococcal sepsis (Infections and infestations) | 2 (2) | 2 (2) | 2 (2) | 2 (2)
Subcutaneous abscess (Infections and infestations) | 9 (9) | 7 (7) | 2 (2) | 3 (3)
Superinfection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Taeniasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tinea capitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 2 (2) | 3 (3) | 3 (3) | 0 (0)
Toxic shock syndrome (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tracheobronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Trichiniasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tuberculosis (Infections and infestations) | 9 (9) | 6 (6) | 6 (6) | 3 (3)
Typhoid fever (Infections and infestations) | 2 (3) | 1 (1) | 3 (3) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 68 (74) | 50 (52) | 43 (45) | 24 (24)
Urinary tract infection (Infections and infestations) | 45 (47) | 26 (28) | 28 (29) | 22 (23)
Urinary tract infection bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection pseudomonal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vaginal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Varicella (Infections and infestations) | 1 (1) | 3 (3) | 1 (1) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Wound sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Accidental exposure to product (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Accidental poisoning (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthropod sting (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchitis chemical (Injury, poisoning and procedural complications) | 4 (4) | 0 (0) | 2 (2) | 0 (0)
Burns first degree (Injury, poisoning and procedural complications) | 4 (4) | 2 (2) | 1 (1) | 1 (1)
Burns second degree (Injury, poisoning and procedural complications) | 6 (6) | 5 (5) | 2 (2) | 3 (3)
Chemical injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chemical poisoning (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 7 (7) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Crush injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Disinfectant poisoning (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dislocation of vertebra (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Exposure to toxic agent (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 3 (3) | 4 (4) | 1 (1) | 2 (2)
Foreign body (Injury, poisoning and procedural complications) | 5 (5) | 0 (0) | 0 (0) | 0 (0)
Foreign body aspiration (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Fractured skull depressed (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Greenstick fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 2 (2) | 4 (4) | 1 (1) | 0 (0)
Herbal toxicity (Injury, poisoning and procedural complications) | 5 (5) | 2 (2) | 2 (2) | 3 (3)
Human bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Limb traumatic amputation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Penis injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Petroleum distillate poisoning (Injury, poisoning and procedural complications) | 4 (4) | 1 (1) | 4 (4) | 1 (1)
Pneumonitis chemical (Injury, poisoning and procedural complications) | 5 (5) | 4 (4) | 4 (4) | 0 (0)
Poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pulmonary contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Sciatic nerve injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Snake bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Soft tissue injury (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 0 (0) | 3 (3)
Thermal burn (Injury, poisoning and procedural complications) | 25 (26) | 24 (24) | 15 (15) | 11 (11)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Vaccination failure (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Wound (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 20 (21) | 6 (6) | 18 (20) | 3 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypoproteinaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Kwashiorkor (Metabolism and nutrition disorders) | 15 (18) | 16 (17) | 17 (17) | 4 (4)
Malnutrition (Metabolism and nutrition disorders) | 54 (58) | 50 (58) | 21 (25) | 19 (21)
Marasmus (Metabolism and nutrition disorders) | 14 (14) | 11 (11) | 4 (4) | 7 (8)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Underweight (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dactylitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rickets (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Torticollis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Acute promyelocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Inflammatory pseudotumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Langerhans' cell histiocytosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arachnoid cyst (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebellar ataxia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebral atrophy (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 102 (122) | 78 (98) | 58 (64) | 32 (45)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Encephalomalacia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 13 (14) | 3 (5) | 2 (2) | 0 (0)
Febrile convulsion (Nervous system disorders) | 344 (466) | 191 (248) | 166 (221) | 103 (127)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hemiparesis (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hemiplegia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Hydrocephalus (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Meningism (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Mental retardation (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metabolic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Monoparesis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myoclonus (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Paraparesis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Speech disorder developmental (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Uraemic encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neurodevelopmental disorder (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Glomerulonephritis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Glomerulonephritis acute (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nephritis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nephrotic syndrome (Renal and urinary disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal tubular necrosis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acquired phimosis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Apnoeic attack (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 15 (21) | 9 (9) | 8 (19) | 7 (7)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 8 (8) | 3 (3) | 5 (7)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 4 (4) | 6 (6) | 4 (4)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Stevens-johnson syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Vitiligo (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Child abuse (Social circumstances) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sexual abuse (Social circumstances) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypovolaemic shock (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Shock (Vascular disorders) | 3 (3) | 3 (3) | 5 (5) | 4 (4)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK257049 [5-17M] Group (N=1479) | GSK257049 [6-12W] Group (N=1462) | VeroRab Comparator [5-17M] Group (N=721) | Menjugate Comparator [6-12W] Group (N=738)
Diarrhoea (Gastrointestinal disorders) | 196 (226) | 0 (0) | 92 (107) | 0 (0)
Enteritis (Gastrointestinal disorders) | 136 (148) | 149 (195) | 65 (74) | 80 (97)
Pain (General disorders) | 493 (688) | 729 (1251) | 132 (165) | 348 (571)
Pyrexia (General disorders) | 1028 (1971) | 966 (1852) | 306 (416) | 408 (660)
Swelling (General disorders) | 352 (491) | 456 (713) | 138 (192) | 272 (407)
Bronchitis (Infections and infestations) | 83 (92) | 69 (80) | 37 (41) | 33 (36)
Conjunctivitis (Infections and infestations) | 126 (135) | 139 (147) | 74 (77) | 81 (87)
Gastroenteritis (Infections and infestations) | 368 (435) | 257 (339) | 159 (188) | 150 (207)
Malaria (Infections and infestations) | 305 (422) | 199 (249) | 207 (289) | 108 (141)
Otitis media (Infections and infestations) | 0 (0) | 73 (82) | 0 (0) | 41 (42)
Pneumonia (Infections and infestations) | 175 (200) | 87 (94) | 72 (84) | 33 (36)
Rhinitis (Infections and infestations) | 123 (139) | 166 (183) | 52 (59) | 94 (109)
Upper respiratory tract infection (Infections and infestations) | 683 (1006) | 655 (1014) | 343 (493) | 344 (503)
Viral upper respiratory tract infection (Infections and infestations) | 111 (126) | 90 (111) | 60 (69) | 49 (55)
Decreased appetite (Metabolism and nutrition disorders) | 444 (609) | 281 (412) | 151 (190) | 114 (158)
Somnolence (Nervous system disorders) | 272 (364) | 302 (475) | 87 (115) | 131 (179)
Irritability (Psychiatric disorders) | 412 (583) | 589 (1017) | 106 (131) | 255 (411)
Cough (Respiratory, thoracic and mediastinal disorders) | 119 (126) | 0 (0) | 47 (54) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 147 (162) | 307 (436) | 57 (66) | 172 (254)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.